#### CLINICAL RESEARCH PROJECT

#### PROTOCOL #11-H-0064

**Drug Name:** aerosolized cyclosporine A in solution with

propylene glycol (CIS) **IND Number:** 109,707

Sponsor: Richard Childs, MD

**Title**: Extension Study (extended access) of Cyclosporine Inhalation Solution (CIS) in lung transplant and hematopoietic stem cell transplant recipients for the treatment of Bronchiolitis Obliterans

Other identifying words: Lung transplant, Single lung transplant, Double lung transplant, Peripheral blood stem cell transplant, Bronchiolitis obliterans syndrome, myeloablative stem cell transplant, nonmyeloablative stem cell transplant, inhaled cyclosporine

# **Principal Investigator:**

| *Nicole Gormley, MD, NHLBI, OCD (V) | 240-402-0210 | WO22 RM2113, FDA, |
|---|---|---|
| | 10903 New Hampshire Ave, Si | lver Spring, MD 20903 |

## **Medically Responsible Investigator:**

| *Richard W. Childs, MD, NHLBI, HB (E) 594-8008 Bldg 10, 0 | 0, CRC 3-5332 |
|-----------------------------------------------------------|---------------|
|-----------------------------------------------------------|---------------|

# **Lead Associate Investigator**

| *Anthony Suffredini, MD, CC, CCMD (E) | 402-3485 Bldg 10, 2C145 |
|----------------------------------------|--------------------------|
| *Anthony Silitredini Will ( ( William) | 4U/-34X3 BIOG III /L 143 |
| minion y bullicum, wib, cc, ccivib (b) | 702-3703 Diag 10, 20173 |

# **Associate Investigators:**

| Clara Chen, MD, CC, Nuclear Medicine (E) | 496-5675 | Bldg 10, 1C401 |
|---|---|---|
| Corina Millo, MD, CC, PET (E) | 402-4297 | Bldg 10, 1C490 |
| Robert Danner, MD, CC, Critical Care (E) | 496-9320 | Bldg 10, 2C145 |
| Sandra Mitchell, PhD, CRNP, AOCN, NCI (E) | 240-276-6929 | Bldg9609, 3E448 |
| Lisa Cook, RN, Research Nurse, HB, NHLBI (E) | 402-5609 | Bldg 10, CRC 3-3485 |
| Tatyana Worthy, RN, HB, NHLBI (E) | 594-8013 | Bldg 10, CRC 3-3485 |
| Nancy Geller, PhD, Director, OBR, NHLBI (E) | 435-0434 | Rockledge 2, 9202 |
| Xin Tian, PhD, Biostatistician, OBR, NHLBI (E) | 435-1298 | RKL2, 9208 |
| Thomas Hughes, PharmD, CC, Pharmacy (E) | 451-0495 | Bldg 10, 1N257 |
| Debra Reda, RN, CC (E) | 496-9320 | Bldg 10, 2C145 |
| Robert Reger, NHLBI (E) | 594-8004 | Bldg 10, CRC 3-5332 |
| Brian Wells, HB, NHLBI (E) | 451-7128 | Bldg 10, 3-1341 |
| Georg Aue, MD, HB, NHLBI (E) | 451-7141 | Bldg 10, CRC 3-3216 |
| * - Investigators who can obtain informed consent | | |

<sup>\* =</sup> Investigators who can obtain informed consent

## **Collaborators:**

Aldo T. Iacono, M.D., Medical Director, Lung Transplant Program U of Md Med Center, 655 West Baltimore Street, Baltimore, Maryland 21201-1559, aiacono@umm.edu 1-800-373-4111

Michael Terrin, MD, Professor of Epidemiology and Medicine, University of Maryland, University of Maryland School of Medicine, 655 West Baltimore Street, Baltimore, Maryland 21201-1559, <a href="maryland.edu">mterrin@epi.umaryland.edu</a> 410-706-6139.

11-H-0064 Am L

Version Date: 10 May 2019

Timothy Corcoran, PhD, Professor of Medicine and Bioengineering, Pulmonary, Allergy and Critical Care Medicine, University of Pittsburgh, NW 628 UPMC Montefiore, 3459 Fifth Ave, Pittsburgh, PA 15213 <a href="mailto:corcorante@MSX.upmc.edu">corcorante@MSX.upmc.edu</a> 412-647-5473.

Independent Medical Monitor: Stewart Levine, MD NHLBI (E) 402-1448, Bldg 10 6D16

# **Collaborating Pharmaceutical Company:**

APT Pharmaceuticals, Inc., 700 Airport Blvd., Suite 350, Burlingame, CA 94010

| Subject of Study: | <u>Number</u> | <u>Sex</u> | <u>Age range</u> |
|---|---|---|---|
| Hematopoietic stem cell transplant recipients (group A | A) 39 | Either | 10-80 |
| Lung transplant recipients (Group B) | 39 | either | 10-80 |
| (No longer enrolling) | | | |
| Total subjects | 78 | either | 10-80 |
| Project involves ionizing radiation? Yes | | | |
| Off site project? | | | |
| Multi-institutional project? No | | | |
| DSMB involved Yes | | | |

11-H-0064 Am L


#### **Precis**

Bronchiolitis Obliterans (BO) is an obstructive lung disease that can affect individuals that have undergone a lung or hematopoietic stem cell transplant. BO has been studied most extensively in lung transplant recipients, where it is considered to represent chronic lung rejection. It is the leading cause of death after lung transplant, with mortality rates up to 55%. In hematopoietic stem cell transplantation, BO is thought to be a manifestation of chronic graft-vs-host disease (GVHD). Up to 45% of patients undergoing hematopoietic stem cell transplantation at the NHLBI develop a decline in pulmonary function. Conventional therapy for patients who develop BO consists of augmentation of systemic immunosuppressants. Systemic immunosuppression has limited efficacy for BO and is associated with deleterious consequences including increased risk of infections and decreased graft-versus tumor/leukemia effects.

Recently, cyclosporine inhalation solution (CIS) in solution with propylene glycol has been shown to improve overall survival and chronic rejection-free survival in lung transplant patients. These findings suggest targeted delivery of immunosuppressive therapy to the diseased organ warrants further investigation as this may minimize the morbidity associated with systemic immunosuppression. However, there currently exists limited data regarding the overall efficacy of inhaled cyclosporine to treat established BO following lung transplantation. Furthermore, inhaled cyclosporine has not been studied in the treatment of BO following hematopoietic stem cell transplantation.

Here, we propose to evaluate the long-term safety and efficacy, of inhaled CIS for the treatment of BO. Enrollment will be offered to subjects who have completed the end of study (week 18 visit) for the initial protocol (Phase II Trial of CIS in lung transplant and hematopoietic stem cell transplant recipients for treatment of Bronchiolitis Obliterans) and who have shown evidence of benefit (either an improvement or stabilization) in BO/BOS with CIS treatment.

Clinical parameters, including pulmonary function tests, will be measured in addition to laboratory markers of the anti-inflammatory response to CIS. Adverse events associated with extended treatment with CIS will be recorded.

*The primary objective* is to provide long-term safety and efficacy data for the use of CIS in hematopoietic transplant patients and lung transplant patients with established BO.

Secondary objectives include investigation of the inflammatory pathways that lead to chronic BO and ascertainment of the long term anti-inflammatory effects of this CSA preparation ex vivo and in vivo.

*Primary endpoint* is efficacy of extended use CIS for BO/BOS. *Secondary endpoints* include the toxicity profile (adverse events), improvement in high-resolution chest CT images, results of peripheral blood and bronchoalveolar cytokine arrays to assess secondary markers of inflammation, and functional capacity measurements using a six-minute walk test.

11-H-0064 Am L Version Date: 10 May 2019

# TABLE OF CONTNETS

- 1. Objectives
- 2. Background
- 3. The investigational product: Inhaled CsA
- 4. Study Design
- 5. Eligibility Assessment
- 6. Treatment Plan
- 7. Study Assessments
- 8. Assessment tools and procedures
- 9. Ancillary Laboratory Research Studies
- 10. Biostatistical Considerations
- 11. Data and Safety Monitoring Plan
- 12. Adverse Events
- 13. Human Subjects Protection
- 14. Pharmaceuticals
- 15. Role of Collaborators
- 16. References

# Appendix

- A MEDWATCH Form FDA 3500A
- B IRB Approved List of Laboratory Research Studies v. 2/5/2013
- C Protocol definitions.
- D Event Characterization and Reporting to the IRB, Clinical Director (CD), and (as applicable) Sponsor

# See Also: PATIENT ASSESSMENT FORMS

- Initial assessment
- Interim clinical assessment
- Human Activity Profile (HAP)
- 6 minute walk
- SF36

11-H-0064~Am~L


#### 1.0 OBJECTIVES

# 1.1 Primary objective:

To provide long-term safety and efficacy data for the use CIS in hematopoietic transplant patients and lung transplant patients with established BO have shown evidence for a benefit with CIS. <u>As of March 2017</u>, lung transplant patients are no longer being enrolled on this protocol.

# 1.2 Secondary Objectives

- To investigate the inflammatory pathways that lead to chronic BO
- To ascertain the long term anti-inflammatory effects of this CSA preparation ex vivo and in vivo

#### 2.0 BACKGROUND

#### 2.1 Introduction

After the first year post lung transplant, BO is the leading cause of death, accounting for 26% of all deaths between post transplant years 1 and 3<sup>(1)</sup>. Annually, approximately 15,000 allogeneic hematopoietic stem cell transplants are performed. BO as a manifestation of chronic graft-vs-host disease (GVHD) can also occur after hematopoietic stem cell transplantation. Up to 45% of patients undergoing hematopoietic stem cell transplantation at the NHLBI develop a decline in pulmonary function, with a significant proportion of these patients being diagnosed with BO <sup>(2)</sup>. Although similarities and differences in the pathogenesis of BO following lung and hematopoietic stem cell transplantation have not been well characterized, both present with similar clinical manifestations and are treated similarly with increased doses of systemic immunosuppressants. The current treatment for BO is inadequate and involves increasing systemic immunosuppression or immune-modulating therapies, which are of marginal efficacy.

## 2.2 Hematopoietic Transplant and BO / BOS

Hematopoietic stem cell transplant is an established therapy for the treatment of many lifethreatening diseases. However, there are many life-long complications associated with this treatment, especially lung disease. Pulmonary dysfunction after hematopoietic stem cell transplant has been well documented, and is one of the most frequent complications seen after transplant (2, 3, 4). The incidence of BO after hematopoietic transplant has been estimated between 5 and 60% (4, 10). The underlying pathophysiology is not completely understood, but it is thought that BO represents a form of chronic GVHD, with the lung epithelium serving as a target for immune-mediated injury induced by transplanted donor T lymphocytes (5). In concert with this proposed mechanism is the observation that GVHD is the greatest risk factor for the development of BO after stem cell transplant (4). This is also supported by the very low incidence of BO occurring after autologous stem cell transplant. It has been proposed that additional factors may have a role in the development of BO. Other factors may include recurrent aspiration due to GVHD induced esophagitis, infection, HLA mismatched transplant, use of busulfan or methotrexate, or lung disease prior to transplant (3, 4).

# 2.3 Lung transplant and BO / BOS

Bronchiolitis obliterans is the characteristic lesion seen on histology in chronic rejection after lung transplant. It is estimated that 50% of lung transplant recipients will develop BOS within five years of transplantation, with mortality rates upwards of 55% (10,8). The pathogenesis of BOS development after lung transplant is thought to have immune and non-immune facets. It has been postulated that

11-H-0064 Am L


airway inflammation and epithelial cell injury result in a disordered repair process that leads to the fibroproliferative obstruction of the small airways. The initial injury may result from allo-immune or immune-independent factors or both, but have a common final pathway, BO. Various immune mediated risk factors, which have been proposed as inciting events include: increased HLA mismatching, acute rejection, and lymphocytic bronchitis and bronchiolitis in the absence of infection. Non-immune mediated risk factors include chronic aspiration, infection, especially with CMV, and ischemic graft injury <sup>(6,10)</sup>.

# 2.4 BO clinical findings and diagnosis

BO is an obstructive lung disease of the small airways. Patients may present with cough, dyspnea, wheezing, or may be asymptomatic at the time of diagnosis. Cough is present in 60-100% of patients and dyspnea in 50-70% <sup>(3)</sup>. In patients who have received a hematopoietic stem cell transplant, signs and symptoms of chronic graft versus host disease (GVHD) affecting other organs are often present.

The gold standard for the diagnosis of BO is histologic. On histology, there is fibrous proliferation affecting the small airways due to injury and inflammation of the epithelial cells. However, histologic evidence of disease is often difficult to obtain due to the patchy nature of the small airway involvement. As such, a set of clinical diagnostic criteria has been proposed by the NIH working group <sup>(7)</sup>. When histology is not available, the term Bronchiolitis Obliterans Syndrome (BOS) is used. The diagnostic criteria for bronchiolitis obliterans syndrome is largely based on the presence of obstructive pattern pulmonary function tests with exclusion of other causes of airway obstruction such as asthma, infection or emphysema.

Criteria for the diagnosis of BOS, as proposed by the NIH working group, are met when all of the following are met:

- FEV<sub>1</sub>/FVC less than 0.7 and a FEV<sub>1</sub> less than 75% predicted
- Evidence of air trapping on high-resolution chest CT or residual volume ≥120%
- Absence of infection in the respiratory tract
- One or more manifestations of chronic GVHD in another organ system
- a 10% decline from pre-transplant baseline in the FEV<sub>1</sub> and one of the following: FEV1/FVC less than 0.7, evidence of air trapping on CT or residual volume ≥120%

It is generally thought that this definition is too restrictive, and it has on more than one occasion excluded patients with biopsy proven BO. As such, in this study we will require for diagnosis of BOS an FEV<sub>1</sub> less than 75% predicted, absence of infection or other causative etiology, a 10% decline from pre-transplant baseline in the FEV<sub>1</sub> and one of the following: FEV1/FVC less than 0.7, evidence of air trapping on CT or residual volume  $\geq$ 120%, or in hematopoietic transplant recipients at least one other manifestation of cGVHD involving another organ system. In lung transplant recipients, the same criteria will be used, but the FEV<sub>1</sub> decline required will be greater than 20% compared to best post-transplant measurement.

#### 2.5 Current Treatment for BO

Current treatment for BO is inadequate and involves increasing systemic immunosuppression or immune-modulating therapies. In patients who are not already on immunosuppressive therapy, as may be the case in hematopoietic stem cell patients, prednisone is commonly used as an initial treatment. If there is no improvement, immunosuppression with cyclosporine or azathioprine is

11-H-0064 Am L


initiated. While on immunosuppression, prophylaxis for pneumocystis carinii and streptococcus pneumonia should be given <sup>(3)</sup>. Despite these treatments, improvement or stabilization in lung function is noted in only 10-60% of patients <sup>(3, 4, 11)</sup>. Additionally, increased immunosuppression is associated with increased risk of infection, morbidity, and disease relapse.

# 2.6 The Investigational Product: Cyclosporine Inhalation Solution

## 2.6.1 Background

Cyclosporine Inhalation Solution (cyclosporine A in solution with propylene glycol, CIS) is a novel therapeutic agent in late stage development designed to deliver cyclosporine topically to the airways of lung transplant recipients in combination with standard immunosuppressive regimens. By administering cyclosporine through an inhaled route, augmented immunosuppression is provided directly to the diseased, target tissue while minimizing the systemic exposure and subsequent toxicity of the parent compound.

# 2.6.2 Pharmacology

CIS consists of the active ingredient cyclosporine (USP) dissolved in propylene glycol. Cyclosporine is among the most common immunosuppressants used for the prevention and treatment of renal, liver, and heart allograft rejection. Cyclosporine has also been demonstrated to extend the graft survival of bone marrow, skin, small intestine, pancreatic, and lung transplants, as well as treat a variety of rheumatologic conditions. Cyclosporine suppresses the immune response by inhibiting evolutionarily conserved signal transduction pathways necessary for T lymphocyte activation and proliferation.

Cyclosporine is an 11 amino acid cyclic peptide derived from a naturally occurring fungus. It is highly lipophilic and can readily cross the cell membrane of T-lymphocytes without receptor activation. Once in the cytoplasm, cyclosporine forms a drug-protein complex with a specific immunophilin (cyclophilin) that can block the function of calcineurin, a T cell serine threonine phosphatase. When blocked, calcineurin cannot facilitate the translocation of a nuclear transcription activation factor (NFAT) from the cytoplasm to the nucleus where it would normally activate transcription of interleukin-2 (IL-2) and other cytokines. As a result, early T cell activation and proliferation are inhibited in a potent manner. By delivering cyclosporine directly to the affected airways, early lymphocyte activation is diminished and intra-graft immune events that can contribute to the development of BO are controlled.

In vivo preclinical pharmacology and pharmacokinetic experiments have not been performed with the current formulation of cyclosporine dissolved in propylene glycol. However, earlier experiments in dogs and rats conducted with cyclosporine dissolved in ethanol revealed that exposure to inhaled cyclosporine was well tolerated and resulted in lung concentrations that were several hundred-fold higher than concentrations in liver, kidney, heart and blood (12). In rat lung transplant models, treatment with inhaled cyclosporine provided protection from allograft rejection compared to untreated animals and led to a dose-dependent reduction in pro-inflammatory cytokine production. Furthermore, the degree of protection was superior to animals treated with cyclosporine via a systemic intramuscular route (13). Similar results were found when inhaled cyclosporine was evaluated in a canine orthotopic lung transplant model (14).

#### 2.6.3 Animal models

11-H-0064~Am~L


Two 28-day inhalational toxicology studies sponsored by Chiron Corporation (Battelle studies N103752 in rats and N103751 in dogs), provide the core data for direct toxicity evaluation (both systemic and local) of both CIS and propylene glycol. These studies were performed with daily dosing at maximally tolerated (rats) or maximally feasible (dogs) doses of CIS. Exposure in these studies was in excess of the maximum clinical exposure, both in terms of overall dose given per day for both cyclosporine and propylene glycol as well as in frequency of dosing (daily in animals vs. three times/week clinically). These studies demonstrated that the local effects of cyclosporine in the respiratory tract should be tolerable in humans at the proposed clinical doses. There was no unexpected systemic toxicity or significant local respiratory system toxicity associated with inhalation exposures up to approximately 2.7 times the maximum human exposure per dose. Mortality associated with the pulmonary effects of CIS was observed in rats at pulmonary deposited doses more than 5 times the maximum human exposure per dose.

Toxicokinetic data generated in these animal studies indicate that after inhalation, lung exposure to cyclosporine is 10 to 20-fold greater than systemic exposure as measured by peak concentrations, trough concentrations, and area under the curve (AUC) analyses. Cyclosporine from the propylene glycol formulation is partially absorbed systemically and does not accumulate with daily repeated dosing. Half-life ( $t_{1/2}$ ) in the blood was consistent with that observed with intravenous (IV) exposure in both rats and dogs. Thus, once the compound reaches the systemic circulation, the disposition should be similar to the disposition of the compound after IV and/or oral administration.

## 2.6.4 Previous Human Experience

The systemic toxicity of cyclosporine has been well characterized in humans and animals. The most common toxicities associated with systemic exposures include renal dysfunction, hypertension, dyslipidemia, hirsutism, headache, increased risk of infections, and tremor. Additional, less common toxicities include gum hyperplasia, hyperkalemia, thrombocytopenia, and seizure. Hypertension, dyslipidemia, and renal dysfunction are particularly prevalent in the lung transplant population with extended use.

As cyclosporine is partially systemically absorbed following inhalation, the risk of systemic toxicities in addition to the risk of local respiratory tract toxicities was evaluated in repeat dose animal studies. After demonstrating efficacy in preclinical canine and rodent transplant models, ethanol-based inhaled cyclosporine was tested in a series of open-label protocols evaluating its safety and efficacy in lung transplant recipients with established BO and/or refractory acute rejection (AR). In patients with established BO, the administration of inhaled cyclosporine in conjunction with standard immunosuppressive therapy led to improvement in rejection histology, stabilization of pulmonary function, and improvement in survival compared to contemporary and historical controls (15,16). In patients with AR that failed to respond to high-dose pulsed methylprednisolone, the administration of inhaled cyclosporine in conjunction with standard immunosuppressive therapy led to improvement in AR histology, improvement in pulmonary function, a decline in pro-inflammatory cytokine production in bronchoalveolar samples, and improvement in survival compared to contemporary control patients (17,18,19). Although these studies demonstrated the safety of inhaled cyclosporine, the ethanol solvent was associated with substantial respiratory tract irritation and was subsequently changed to propylene glycol.

These open label protocols were followed by a randomized, double-blind, placebo-controlled study of CIS designed to test the efficacy of CIS in preventing lung allograft rejection and improving outcomes when given as prophylactic therapy (8). A total of 56 patients were enrolled within 7 to 42 days following their single- or double-lung transplant and treated with either CIS or placebo

11-H-0064 Am L Version Date: 10 May 2019

(propylene glycol alone). Of these 56 patients, a total of 26 patients received CIS and 30 patients received placebo. All patients underwent an initial dose-titration period to find the maximum tolerated dose up to a protocol-specified maximum of 300 mg (or the equivalent volume of propylene glycol in the placebo group). After this 10-day period, patients were to continue therapy 3 times per week for a period of 2 years. The study concluded on August 21, 2003, when the 56th patient completed the full 2 years of treatment. Follow-up in the randomized cohort ranged from 24 to 56 months.

Results of the study demonstrated that treatment with CIS was associated with a 79% decreased risk of death compared with treatment with placebo (hazard ratio [HR] = 0.213; log-rank p = 0.007). This statistically significant survival advantage was also observed when stratified by transplant type, primary diagnosis, cytomegalovirus (CMV) donor positive/recipient negative mismatch, or the occurrence of a grade 2 or higher AR episode prior to enrollment. The survival advantage from CIS treatment may have arisen from a decreased incidence of chronic rejection, consistent with the mode of delivery to the airway epithelium. Patients treated with CIS had significantly improved chronic rejection-free survival (HR = 0.28; log-rank p = .001) compared with patients treated with placebo. Chronic rejection was diagnosed either through biopsy by the presence of BO or clinically by the presence of bronchiolitis obliterans syndrome (BOS). Among the 30 placebo-treated patients, only 8 (27%) survived free of chronic rejection compared with 18 (69%) CIS-treated patients. Analyses of BOS-free survival and BO-free survival revealed comparable results. However, treatment with CIS did not lead to significant difference in the occurrence of AR (p = 0.73).

Further analysis of the study population revealed that CIS had a favorable safety profile, and long-term administration did not lead to exacerbations of known toxicities of oral and intravenous cyclosporine. In particular, there was no evidence that administration of CIS led to increased risk of nephrotoxicity, neurotoxicity, increased risk of infections, or increased risk of malignancies. Treatment with CIS was found to be associated with respiratory tract irritation and bronchospasm, but these events were generally mild/moderate, occurred early in patients' treatment course, diminished with time, and were not associated with the development of more serious respiratory complications. These findings were consistent with the analysis of the larger 70 patient safety database.

In March 2005, an open label early access treatment IND was initiated. The purpose of this protocol was to provide CIS to lung transplant physicians for use in suitable lung transplant recipients. Since that time, over 60 lung transplant recipients have received CIS. Data collection is limited to early tolerability subject diaries and serious adverse events (SAEs). Analysis of this safety database has not led to the emergence of any new safety findings. However, in recipients with poor pulmonary reserve (such as those with advanced BOS), intolerance to dosing is more common, and dose titration to the maximal 300 mg dose is sometimes not possible.

The safety and efficacy of CIS in preventing chronic rejection and improving survival in this population of lung transplant patients has been previously demonstrated in a randomized double-blind, placebo-controlled, clinical study. This study was the basis for a new drug application (NDA) to regulatory authorities. This application received an approvable letter, with approval contingent on additional supporting clinical data. There is currently a multicenter, phase III, randomized, controlled trial designed to assess the efficacy of prophylactic inhaled cyclosporine for the prevention of bronchiolitis obliterans in lung transplant recipients. However, there currently exists limited data on the efficacy of CIS in propylene glycol to treat established BO/BOS occurring in lung transplant recipients and no data in HSCT recipients with established BOS.

11-H-0064 Am L Version Date: 10 May 2019 PI: N. Gormley

## 2.7 Rational for Dose, Route and Schedule

Because patients who are eligible for this trial have already demonstrated a clinical response to CIS, continuation of therapy is warranted. Patients will be continued on their individualized maximum tolerated dose from the prior study.

Previous clinical trials have taken place at the University of Pittsburgh Medical Center (UPMC), which is a leading center in lung transplantation research and clinical management of lung transplant recipients. We will conduct this study using the same dose of CIS as was used in the Pittsburgh chronic lung rejection prevention trial, specifically 300 mg cyclosporine (or maximally tolerated dose up to 300 mg) administered three times per week. The formulation is 325 mg cyclosporine in 5.2 mL of propylene glycol (62.5 mg/mL) (150 mg to 300 mg inhalation dose, total volume 2.4 to 4.8 ml).

# 2.8 Rationale for including pediatric patients

There are no alternative treatment options for children who develop this often, fatal consequence of lung or hematopoietic stem cell transplantation. Therefore, the potential efficacy of extended therapy with inhaled CsA would be relevant to children. Again, only those patients that have demonstrated a response to CIS will be eligible for enrollment in this long-term protocol. At present there is no data on the long-term use of CIS in children. However, studies investigating inhaled medications in children vs. adults suggest systemic absorption of inhaled drugs, even when administered at the same doses, are not higher in pediatric populations compared to adults. A study investigating lung deposition of inhaled steroids in children and adults (children 2-3 years, children 4-6 years, adults 10-41 years) with asthma receiving the same fixed dose of inhaled budesonide (2 x 200 ug via Nebuchamber pMDI with mouthpiece and nose clip) showed that systemic absorption of budesonide (as measured by plasma AUC) was similar for all age groups<sup>21</sup>. This data suggests, from a safety standpoint, that the prescribed dose of inhaled budesonide need not be adjusted for age. A previous pharmacokinetic study of CIS in adults with BO/BOS found that the systemic exposure of CSA using comparable doses of CIS as used in this study, is about 7-fold lower than is achieved with CSA given orally (Neoral®) at comparable doses<sup>22</sup>. Maximum blood concentrations of cyclosporine after aerosol administration of CIS ranged from 119 to 402 ng/mL, while 24 hr concentrations ranged from 9 to 48 ng/mL (versus reported C<sub>max</sub> concentrations of 1555 ng/mL and trough concentrations of 268 ng/mL in liver transplant recipients, according to the Neoral® label). From these data we infer that inhaled CIS in pediatric populations age 10 and older will not result in toxic systemic levels of CSA however adjustments will be made for pediatric dosing per APT recommendations. We will closely monitor their plasma cyclosporine levels during the study.

## 2.9 Rationale for pediatric dosing

(per Charles Johnson, MD, Chief Medical Officer, APT Pharmaceuticals)

The main safety concerns in this age group are to ensure that there is not excessive systemic exposure to cyclosporine and there is no impact on lung function. It is normal practice to dose the currently licensed forms of cyclosporine (eg Neoral) on the basis of weight and monitor blood levels of cyclosporine. In addition, data from Chua et al, 1994 in 8 children (median age 10.8 y) with cystic fibrosis showed that in this age group, age was not a factor in the amount of drug deposited following aerosol delivery. Therefore, it is proposed to use weight as the main determinant of dose and divide the pediatric population into two groups on the basis of weight. Current experience in the adult population indicates that six adult subjects weighing less than 45 Kg (range 34.5 - 44.3 Kg) have been exposed to CIS. All six achieved a dose of 300 mg in the titration phase and none have reported

 $11\text{-H-}0064\;Am\;L$ 


adverse events associated with study drug. The lightest subject had a peak serum cyclosporine level of 39.7 ng/mL one hour after the inhalation. This level is substantially below the therapeutic level set for systemic therapy (250 -350 ng/mL), suggesting that systemic exposure is not likely to be dose limiting at least in children above 35 kg.

Since the same nebulizer/compressor system will be used in the pediatric population, the proportion of nominal dose which is emitted at the mouth-piece will remain constant. The lung delivered dose is then dependent upon minute ventilation (slightly lower than adults across this age group) and air entrainment (less dilution of the dose due to a lower inspiratory flow rate in children) these factors will exist as a continuum across the population having a greater impact in the smaller younger subjects. Although the adult data suggests that there is a wide therapeutic margin (very low systemic cyclosporine exposure) it would seem prudent to reduce the nominal dose in the youngest, lightest population. The proposed dose for the pediatric age group is as follows:

```
Weight \geq 35 Kg dose at 300 mg
Weight \leq 35 Kg dose at 200 mg
```

This dosing schedule is being used in a multicenter phase III Trial, NCT00755781.

## 2.10 Clinical and Scientific Justification

Because patients who are eligible for this trial have already demonstrated a clinical response to CIS, continuation of therapy is warranted. Therefore, we propose this extended access phase II clinical trial designed to evaluate the safety and efficacy of long term use of inhaled cyclosporine in lung transplant and hematopoietic transplant recipients.

This study also seeks to further define the inflammatory pathways associated with BOS in stem cell transplant and lung transplant recipients and to investigate and compare similarities and differences in the pathogenesis of BOS following long-term therapy. Bronchoalveolar lavage will be studied using multiplex cytokine arrays, flow cytometry, and gene expression profiling. These studies will be performed on samples collected from patients and will promote further delineation of the underlying pathogenesis in BOS. Additionally, this study will examine the anti-inflammatory effects of cyclosporine on mediators of inflammation and differential gene expression in these populations. This has not been thoroughly studied in hematopoietic stem cell transplant recipients. This study evaluating the long term safety and efficacy of aerosolized cyclosporine will contribute to a greater understanding of the pathogenesis of bronchiolitis obliterans, and set the stage for larger trials in hematopoietic stem cell transplant and lung transplant recipients.

## 3.0 INVESTIGATIONAL PRODUCT

Please refer to the Investigator's brochure for Cyclosporine Inhalation Solution (CIS).

#### 4.0 STUDY DESIGN

The study is designed as extended access study following response to initial treatment on the companion non-randomized, Phase II study of aerosolized cyclosporine A in solution with propylene glycol (CIS) in hematopoietic stem cell transplant recipients or lung transplant recipients who have been diagnosed with biopsy proven bronchiolitis obliterans or Bronchiolitis Obliterans Syndrome. As of March 2017 this study is no longer enrolling lung transplant recipients.

 $11\text{-H-}0064\;Am\;L$ 


Improvement FEV1 10%

CSA continued at

maximum tolerated dose,

not to exceed 300mg

Stable
FEV1 <10% increase
or <10% decrease

Continued dosing will be dependent on response and tolerance

Subjects may continue as long as they have clinical benefit.

Tapering will be attempted in patients with stable disease

Maximum of 39
PBSCT and 39 lung
transplant pt who
have completed
10-H-0196

| | | | | | | | | | $\longrightarrow$ |
|---|---|---|---|---|---|---|---|---|---|
| Baseline | Wk 24 | Wk 30 | Wk 36 | Wk 42 | Wk 48 | Wk 54 | Wk 60 | Wk 70 | After |
| (week 18 | | | | | | | | | Wk 70 |
| assessment)<br>PFTs | PFTs | PFTs | PFTs | PFTs | PFTs | PFTs | PFTs | PFTs | PFTs |
| Labs | Labs | Labs | Labs | Labs | Labs | Labs | Labs | Labs | (BAL and CT |
| BAL | | BAL | | BAL | | BAL | | BAL | if indicated) |
| QOL | | СТ | | СТ | | СТ | | QOL | |
| СТ | | | | Progression* | | | | СТ | |
| | | | FEV1≥20% | decline, worse | ning status, | | | | |

<sup>\*</sup> Based on two successive measures at least two weeks apart

11-H-0064 Am L


## 5.0 ELIGIBILITY ASSESSMENT

#### 5.1 Inclusion criteria

- 5.1.1 Completed the End of Study visit (week19) on the initial protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans) in the preceding twelve weeks
- **5.1.2** Patients have shown evidence for a clinical benefit to CIS as evidenced by one or more of the following:
  - **5.1.2.1** Improvement in pulmonary function defined by a 10% or more increase in the FEV<sub>1</sub> at week 18, confirmed with repeat PFTs at least 1 week apart.
  - **5.1.2.2** In patients with progressive disease at study entry on the initial protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans), stabilization in pulmonary function, defined as less than a 10% improvement in FEV<sub>1</sub> or less than 10% decline in FEV<sub>1</sub> at week 18, confirmed with repeat PFTs at least 1 week apart.
  - 5.1.2.3 In patients with stable disease (active BOS stable by FEV1 criteria) at study entry on the initial protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans), stabilization in pulmonary function, defined as less than a 10% improvement in their FEV1 or less than 10% decline in FEV1, and a decrease in the dose of one or more systemic immunosuppressants by at least 20% \*(sustained for 3 weeks, excluding adjustments made for target drug levels)
    \* The criteria for study entry on this extension protocol are not the same as the criteria for response on the primary protocol to allow for entry of patients on this extension protocol, which is deriving some clinical benefit, but have not met the full response

# 5.2 Exclusion criteria

**5.2.1** More than a twelve week gap in study drug administration (CIS)

criteria as defined in the primary protocol.

- **5.2.2** Evidence of uncontrolled, pulmonary infection
- **5.2.3** ECOG performance status greater than or equal to 3
- **5.2.4** Patient pregnant or breast feeding or not willing to continue the use of an approved method of birth control
- **5.2.5** Life expectancy less than 18 weeks
- **5.2.6** History of hypersensitivity reaction to propylene glycol
- **5.2.7** Documented allergy or intolerance to CIS

11-H-0064 Am L


- **5.2.8** History of untreated coronary insufficiency, severe cardiac arrhythmias, and/or uncontrolled hypertension.
- **5.2.9** Serum creatinine >2.5 mg/dl
- **5.2.10** Inability to comprehend the investigational nature of the study and provide informed consent

#### 6.0 TREATMENT PLAN

## 6.1 Pre-treatment Medication (albuterol)

Subjects will receive metered dose inhaler albuterol, 2 puffs as needed for prevention of bronchospasm or 3 ml solution for nebulization. Patients may receive levalbuterol in place of albuterol or not receive pre-treatment.

- **6.1.1 Inhalation device:** Subjects will be instructed regarding the use of the inhalation device as follows:
  - Shake the inhaler well.
  - Breathe out as completely as possible through your mouth.
  - Hold the canister with the mouthpiece on the bottom, facing you and the canister pointing upward. Place the open end of the mouthpiece into your mouth. Close your lips tightly around the mouthpiece.
  - Breathe in slowly and deeply through the mouthpiece. At the same time, press down once on the container to spray the medication into your mouth.
  - Try to hold your breath for 10 seconds, remove the inhaler, and breathe out slowly.
  - Wait 10 minutes before beginning cyclosporine nebulizer treatment.
- **6.1.2 Nebulizer:** Subjects will be instructed regarding the use of the nebulizer device as follows:
  - Before treatment, wash your hands with soap and water and dry completely.
  - Place the air compressor on a sturdy surface that will support its weight. Plug the cord from the compressor into a properly grounded (three-prong) electrical outlet.
  - Carefully measure medications exactly as you have been instructed and put them into the nebulizer cup.
  - Assemble the nebulizer cup and mask or mouthpiece.
  - Connect the tubing to both the aerosol compressor and nebulizer cup (with filter if beginning treatment with cyclosporine).
  - Turn on the compressor to make sure it is working correctly. You should see a light mist coming from the back of the tube opposite the mouthpiece.
  - Sit up straight on a comfortable chair. If the treatment is for your child, he or she may sit on your lap. If you are using a mask, position it comfortably and securely on you or your child's face. If you are using a mouthpiece, place it between you or your child's teeth and seal the lips around it.
  - Take slow, deep breaths.
  - Continue the treatment until the medication is gone (an average of 10 minutes for albuterol). The nebulizer will make a sputtering noise, and the cup will have just a little medication remaining.

 $11\text{-H-}0064\;Am\;L$ 


- If dizziness or jitteriness occurs, stop the treatment and rest for about 5 minutes. Continue the treatment, and try to breathe more slowly. If dizziness or jitteriness continues to be a problem with future treatments, inform your doctor.
- During the treatment, if the medication sticks to the sides of the nebulizer cup, you may shake the cup to loosen the droplets.
- After each treatment, rinse the nebulizer cup thoroughly with warm water, shake off excess water, and let air dry.
- Wait 10 minutes before beginning cyclosporine nebulizer treatment.
- 6.1.3 Concomitant Medications of Concern with albuterol (concurrent use will be per PI discretion and carefully monitored) Subjects will be queried as to what prescription medications, vitamins, nutritional supplements, and herbal products they are taking, or have stopped taking within the past two weeks as medication dose adjustments may be required or subjects carefully monitored for side effects with the following medications:
  - beta blockers such as atenolol (Tenormin), labetalol (Normodyne), metoprolol (Lopressor, Toprol XL), nadolol (Corgard), and propranolol (Inderal); digoxin (Lanoxin); diuretics; epinephrine (Epipen, Primatene Mist); other inhaled medications used to relax the air passages such as metaproterenol (Alupent) and levalbuterol (Xoponex); and medications for colds
  - antidepressants such as amitriptyline (Elavil), amoxapine (Asendin), clomipramine (Anafranil), desipramine (Norpramin), doxepin (Adapin, Sinequan), imipramine (Tofranil), nortriptyline (Aventyl, Pamelor), protriptyline (Vivactil), and trimipramine (Surmontil); and monoamine oxidase (MAO) inhibitors, including isocarboxazid (Marplan), phenelzine (Nardil), selegiline (Eldepryl, Emsam), and tranylcypromine (Parnate).
- **6.1.4** Subjects will also be instructed to discontinue albuterol and notify the research team immediately if they:
  - Become pregnant, plan to become pregnant, or are breast-feeding.
  - Experience severe wheezing and difficulty breathing immediately after it is inhaled.
- 6.1.5 Subjects will be instructed not to administer the albuterol and /or study drug on the day of assessments, as the albuterol and/or CsA may complicate the interpretation of the pulmonary function testing.

## 6.2 Study Drug (Aerosolized Cyclosporine A in solution with Propylene glycol) Administration

## 6.2.1 Treatment plan:

Subjects will continue self administration of aerosolized cyclosporine A in solution with propylene glycol using a Sidestream nebulizer with the Invacare Mobilaire compressor at 30 psi at the maximum tolerated dose established during participation on the initial protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans), 3 times weekly (150 mg to 300 mg inhalation dose, total volume 2.4 to 4.8 ml). Continued dosing will be dependent on response and tolerance.

Hematopoietic stem cell transplants (Group A)

 $11\text{-H-}0064\;Am\;L$ 


- 1. Any patient that has continued improvement in lung function, as defined by 10% or more increase in FEV<sub>1</sub>, as compared to their new baseline FEV<sub>1</sub> value, determined by average of week 18 and 19 PFT assessments on the initial study (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans), and/or continued success with weaning systemic immunosuppressants will be maintained on CIS with no effort to taper CIS.
- 2. Patients who show stabilization in PFTs for 6 months, as defined by less than 10% increase in FEV<sub>1</sub> or less than 10% decline in FEV<sub>1</sub>, as compared to their new baseline FEV<sub>1</sub> value, determined by average of week 18 and 19 PFT assessments on initial treatment study (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans), that are either off systemic immunosuppressants or cannot have further tapering of their systemic immunosuppressants, may undergo tapering of CIS, at the discretion of the PI.
  - a. Patients successfully tapered off CIS will continue to have clinical assessments and PFTs performed at 6 week intervals and will be taken off study should PFTs remain stable (in the absence of a need for increased systemic immunosuppression for BO/BOS) for a period of 12 months off therapy.
  - b. Patients who have worsening of BO/BOS associated with tapering CIS will have the CIS reinitiated at the patient's previously defined maximal tolerated dose.
- 3. Any subject that demonstrates disease progression, as defined by a 20% or more decline in FEV<sub>1</sub> on two successive measurements at least 3 weeks apart, or those who require an increase in the existing dose of one or more immunosuppressive therapies by at least 25% (sustained for 3 weeks, excluding adjustments made for target drug levels) above baseline levels from the primary protocol or the addition of new immunosuppressive therapies (sustained for 3 weeks) due to worsening symptoms related to BO/BOS, will be categorized as a treatment failure and will discontinue study drug administration and proceed with end of study drug assessment.

## Lung transplant recipients (Group B) (No longer enrolling)

- 1. Any patient that has improvement or stabilization of lung function, as measured by PFTs will remain on CIS with no attempts to taper CIS.
- 2. Any subject that demonstrates disease progression, as defined by a 20% or more decline in FEV<sub>1</sub> on two successive measurements at least 3 weeks apart, or those who require an increase in the existing dose of one or more immunosuppressive therapies by at least 25% (sustained for 3 weeks, excluding adjustments made for target drug levels) above baseline levels from the primary protocol or the addition of new immunosuppressive therapies due to worsening symptoms related to BO/BOS, will be categorized as a treatment failure and will discontinue study drug administration and proceed with end of study drug assessment.

**Deviation plan for a missed dose:** Subjects will be treated with CIS three times weekly ideally on Monday, Wednesday, and Friday of the week. Should a subject miss a scheduled dose of CIS, we will attempt to alter the dosing regimen for that week so that the subject will still receive three doses of CIS over a week with a limit of 1 dose per day. Data will be captured and reported for subjects who deviate from the treatment plan.

**Medication Holds:** During study participation, subjects may be instructed to hold administration of CIS for development of an adverse event or other reason at the discretion of the PI. Information pertaining to the reason for and the duration of the medication hold will be captured in the patient's

11-H-0064 Am L Version Date: 10 May 2019

medical record. If study drug is held for more than 7 days, the time of the hold will not be counted towards the overall study week count. Study drug can be held for up to 12 months.

## 6.2.2 Special Instructions Regarding the Administration of Aerosolized Cyclosporine A

Patients will follow nebulizer instructions (section 6.1.2) with the following instructions specific to CsA: Continue the treatment until the medication is gone (approx. 10-30 minutes for cyclosporine).

A new nebulizer should be used after albuterol administration. Aerosolized CsA is provided in single use vials. Any CsA remaining in the vial after administration should be discarded immediately.

Subjects will be given a medication log and asked to record their CIS administration on the log. Subjects will be encouraged to capture this information, but failure to comply with this request will not be reported as a protocol deviation.

## **6.2.3 Permitted Concomitant Medications**

Post Transplant Medications:

Subjects that require an increase in the existing dose of one or more immunosuppressive therapies by at least 25% above baseline levels from the primary protocol due to worsening BOS symptoms (sustained for 3 weeks, excluding adjustments made for target drug levels) or the addition of new immunosuppressive therapies (sustained for 3 weeks) due to worsening symptoms related to BO/BOS, will be considered treatment failures. However, if the increase or addition of new immunosuppressive therapies is for GVHD not involving the lung or is to maintain baseline drug levels, this data will be captured and the patient will continue on study. Efforts will be made to make no changes in existing medical therapies other than tapering immunosuppressants in patients who have PFTs showing stable or improved pulmonary function. Again, this data will be captured.

## Lung Infection Prophylaxis:

Lung infection prophylaxis will be at the discretion of the PI, taking into account the patient's other concomitant medications and medical history. The following are guidelines:

- For PCP pneumonia prophylaxis, subjects will take Bactrim, one double strength tablet (800/160mg) orally three times weekly or aerosolized pentamidine 300mg every four weeks by inhalation.
- For antiviral prophylaxis, subjects will receive acyclovir 800 mg twice daily Pediatric patients less than 40kgs will receive acyclovir 20mg/kg po twice daily to a maximum dose of 800mg twice daily.
- For antibacterial prophylaxis, subjects will receive penicillin 500mg twice daily or for penicillin allergic patients, azithromycin 250mg daily.
- Subjects who are already on adequate, alternative prophylaxis agents prescribed by their primary transplant teams can remain on their prior regimens.

# 6.2.4 Concomitant Medications of Concern with CsA (concurrent use will be per PI discretion and carefully monitored)

11-H-0064 Am L


- Due to potential for drug interactions, other short acting sympathominetic aerosolized bronchodilators, beta-adrenergic receptor blocking agents, digoxin, monoamine oxidase inhibitors or tricyclic antidepressants will be allowed per PI discretion.
- Due to the potential for compromising the primary endpoint, subjects requiring an increase in systemic immunosuppression or who initiate new immunosuppressive agents, such as oral tacrolimus, CSA, prednisone, mycophenolate mofetil (MMF) or azathioprine due to symptoms of GVHD *not* involving the lung, will remain on study and will have concurrent use of these medications carefully tracked and accounted for during and at the end of study data analysis.
- Cyclosporine can interfere with or be affected by multiple drugs due to its metabolism through the CYP3A4 enzyme. As such, patients who are taking medications which, are either substrates for, inducers of, or inhibitors of CYP3A4 (i.e. oral cyclosporine) will be closely monitored (see appendix c).

# 7.0 CLINICAL MONITORING PLAN

Human Biologic materials will be collected as follows for the clinical evaluation and management of the patient. Samples will be ordered and tracked through the CRIS screens. Should a CRIS screen not be available, the NIH form 2803-1 will be completed and will accompany the specimen and be filed in the medical record.

- **7.1 On study assessments:** Subjects will be asked to return to the NIH Clinical Center the end of Week 24, 30, 36, 42, 48, 54, 60 (+/- 7 days) for the following assessments:
  - Interim assessment with emphasis on symptomatology
  - Vital signs
  - ECOG performance status
  - Review of concomitant medications and adherence
  - CBC with differential (when possible, done concurrently with post transplant monitoring)
  - Acute Care, Mineral and Hepatic Panels (when possible done concurrently with post transplant monitoring)
  - Plasma cyclosporine level
  - Peripheral blood samples
  - Repeat Serum Beta- HCG in women of childbearing potential
  - Pulmonary Function tests
    - Forced Spirometry
    - Slow Spirometry
    - o Lung volumes with nitrogen washout
    - o Single Breath Diffusion
    - Six minute walk test
    - o Exhaled Nitric Oxide measurement (in a subset of subjects)
    - o Review of Peak Flow measurements
  - Bronchoscopy and bronchoalveolar lavage (BAL) (Weeks 30, 42, 54 only)\* BAL to be analyzed by
    - o Luminex cytokine arrays
    - o Flow Cytometry
    - Gene expression profiles

 $11\text{-H-}0064\;Am\;L$ 


- o Proliferative, cytotoxic, and apoptotic response of BAL lymphocytes to 3<sup>rd</sup> party epithelial cells and allogeneic lymphocyte population
- T regulatory cell quantification by real time PCR
- High Resolution Chest CT (weeks 30, 42, 54 only)\*

## 7.2 End of week 70 and end of study assessments

Patients will be monitored at week 70 (+/- 1 week) and at end of study participation with the following assessments:

- Assessment with emphasis on symptomatology
- Vital signs
- ECOG performance status
- Review of concomitant medications and compliance
- CBC with differential (if possible, done concurrent with post transplant monitoring)
- Acute Care, Mineral and Hepatic Panels (if possible, done concurrently with post transplant monitoring)
- Plasma cyclosporine level
- Repeat Serum Beta- HCG in women of childbearing potential
- Pulmonary Function tests
  - Forced Spirometry
  - Slow Spirometry
  - o Lung volumes with nitrogen washout
  - Single Breath Diffusion
  - o Six minute walk test
  - o Exhaled Nitric Oxide measurement (in a subset of subjects)
  - o Review Peak Flow measurements
- Bronchoscopy and bronchoalveolar lavage (BAL)\*
  - Luminex cytokine arrays
  - o Flow Cytometry
  - Gene expression profiles
  - o Proliferative, cytotoxic, and apoptotic response of BAL lymphocytes to 3<sup>rd</sup> party epithelial cells and allogeneic lymphocyte population
  - T regulatory cell quantification by real time PCR using primers to fox p3
- Peripheral blood samples
- High Resolution Chest CT\*
- Quality of life assessments
  - o SF36
  - o GVHD questionnaire (PBST transplant patients only)
  - o HAP Questionnaire
  - o CRQ-SAS questionnaire
  - o Comfort of study drug administration

## 7.3 Long term follow up after Week 70 until withdrawal from study

After Week 70 assessments are completed, patients will return to the NIH Clinical Center every 6-12 weeks for routine assessment, physical exam and PFTs. Chest CTs, bronchoscopies and BALs will only be done as clinically indicated. The study drug will be made available until it is

11-H-0064 Am L


<sup>\*</sup> Bronchoscopy and High-resolution CT scans are optional unless clinically indicated.

<sup>\*</sup> Bronchoscopy and High-resolution CT scans are optional unless clinically indicated.

commercially available, or until the pharmaceutical company (APT Pharmaceuticals) withdraws the NDA, or for six months if APT Pharmaceuticals undergoes a change of control.

# 7.4 International and Long-distance Subjects

Patients that are travelling internationally or more than 50 miles away from the NIH, at the discretion of the principal investigator, may have their schedules modified. The week 30 evaluation will be a required assessment. Thereafter, patients may be seen at either 6 week, 12 week, or 24 week intervals depending on the ease of travel, medical support systems at home, and the PIs recommendations. If feasible, some pulmonary function tests and laboratory data may be obtained from home medical facilities.

## 8.0 ASSESSMENT TOOLS and PROCEDURES

Other than the pre-study evaluations to determine eligibility/baseline status and subsequent PFTs used to guide therapy, patients will be able to refuse any radiologic test or bronchoscopy procedure unless clinically indicated.

# 8.1 Pulmonary Function tests

**Spirometry** measures how much and how quickly air is moved in and out of the lungs. For these tests, the subject breathes into a mouthpiece attached to a recording device (spirometer). The information collected by the spirometer may be printed out on a chart called a spirogram. The more common lung function values measured used to assess the subjects on this trial will include:

**Forced vital capacity (FVC)**. This measures the amount of air you can exhale with force after you inhale as deeply as possible.

Forced expiratory volume (FEV). This measures the amount of air you can exhale with force in one breath. The amount of air you exhale may be measured at 1 second (FEV<sub>1</sub>).

**Peak expiratory flow (PEF)**. This measures how quickly you can exhale. It is usually measured at the same time as your forced vital capacity (FVC).

**Total lung capacity (TLC)**. This measures the amount of air in your lungs after you inhale as in your lungs after a normal exhale (FRC) and the amount after you exhale with force (RV).

Maximum voluntary ventilation (MVV). This measures the greatest amount of air you can breathe in and out during one minute.

**Exhaled Nitric Oxide measurement**. This measures the amount of nitric oxide exhaled in your breathe after exhalation. This will be performed in a subset of subjects based on the availability of testing staff and scheduling.

**Lung Volumes using Nitrogen Washout.** This measures the total lung capacity and provides an estimate of residual volume of the lung.

11-H-0064 Am L


**Diffusing Capacity of the lungs for carbon monoxide (DLCO)**. This measures the ability of the lungs to transfer gas from inhaled air to the red blood cells in pulmonary capillaries.

**Peak Flow Measurements:** Patients will be given a home peak flow meter that will measure their peak flow and FEV1. The results will be recorded, and patients will be given a level below which, they should call the research team. Patients with a decline in peak flow of >20% compared to pretreatment baseline will be instructed to return to the NIH for formal pulmonary function testing. Subjects will be encouraged to perform peak flow testing daily, however, failure to perform peak flow measurements will not be considered a protocol deviation.

# 8.2 Bronchoscopy and bronchoalveolar lavage (BAL)

Bronchoalveolar lavage (BAL) is a medical procedure in which a bronchoscope is passed through the mouth or nose into the lungs and fluid is squirted into a small part of the lung and then recollected for examination. A BAL sample (minimal 30 mL) will be obtained from upper and lower lobes using conventional techniques. The following research investigations will be performed: Luminex cytokine arrays, flow Cytometry, gene expression profiles, examination of proliferative, cytotoxic, and apoptotic response of BAL lymphocytes to 3<sup>rd</sup> party epithelial cells and allogeneic lymphocyte population, and T regulatory cell quantification by real time PCR using primers to fox p3.

## 8.3 High Resolution Chest CT

HRCT is performed using a conventional CT scanner. However, imaging parameters are chosen so as to maximize spatial resolution:

- A narrow slice width is used (usually 1-2 mm)
- A high spatial resolution image reconstruction algorithm is used
- Field of view is minimized, so as to minimize the size of each pixel
- Other scan factors (e.g. focal spot) may be optimized for resolution at the expense of scan speed

As HRCT's aim is to assess a generalized lung disease, the test is conventionally performed by taking thin sections 10-40 mm apart. The result is a few images which should be representative of the lungs in general, but which cover only approximately one tenth of the lungs.

Intravenous contrast agents are not used for HRCT as the lung inherently has very high contrast (soft tissue against air).

# 8.4 Six Minute Walk Test

The six-minute walk test is generally used at the start of a Pulmonary Rehabilitation program and/or in the evaluation of lung transplant and will be used in this study to evaluate the primary endpoint, which is change in BO status. The object of this test is to walk on a flat surface such as a hallway for 6 minutes during which time subjects will be asked to rate their degree of breathlessness and fatigue levels. The distance walked during the 6 minutes is measured.

Blood pressure, heart rate, respiratory rate, and resting blood saturation by pulse oximetry will be taken after the test. Oxygen saturation will be taken during the walk. Subjects will be asked to assess their breathing status using a 0-10 scale.

 $11\text{-H-}0064\;Am\;L$ 


## Subjects will be instructed to:

- Wear comfortable clothing
- Wear shoes that are comfortable to walk in, such as tennis shoes.
- Take their medications as prescribed.
- Eat a light meal before early morning or early afternoon tests.
- Not to exercise vigorously within 2 hours of beginning the test.

## 8.5 Quality of Life Measurements

Participants sixteen years and older that speak English will perform self-report questionnaires using the SF36, Human Activity Profile (HAP), Chronic Respiratory Disease Questionnaire Self-Administered Standardized CRQ-SAS), and a GVHD questionnaire. These assessments will occur at the week 70 assessment and at end of study assessment.

- The SF36 is a 36 item self-report questionnaire that measures the impact of physical and emotional health status on functional performance. It has been used extensively, and is accepted by the U.S. Food and Drug Administration as proof of therapeutic benefit for improved functioning and other patient-reported outcomes.
- The HAP is a 94-item questionnaire that assesses the frequency with which individuals perform common activities.
- The CRQ-SAS is a 20-item questionnaire that assesses dyspnea, fatigue, emotional functioning, and mastery.
- A GVHD questionnaire (PBSC transplant patients, group A) designed by Lee and colleagues is a 30-item symptom scale with seven subscales to capture cGVHD symptom burden.

## 9.0 ANCILLARY LABORATORY RESEARCH STUDIES

- **9.1 Sample Collection:** During the course of this study, blood and bronchoalveolar lavage samples will be collected for correlative laboratory research studies.
- 9.2 Intended use: These specimens will not be used for diagnostic purposes. Studies conducted on these samples will not be used in assessing the primary endpoint but are undertaken for secondary endpoints (Tissue pathogenesis of BO as detailed below) and/or exploratory ancillary research, which are approved by the NHLBI IRB and listed in Appendix B of the protocol. As these tests are being performed for secondary or exploratory purposes, failure to obtain the tests will not be considered a protocol deviation.

#### 9.2.1 Multiplex cytokine arrays

Biopsies, BAL, and peripheral blood samples will be prepared for multiplex cytokine array analysis. Multiplex bead arrays allow one to independently and quantitatively assay multiple analytes simultaneously in small volumes of material.

## 9.2.2 Flow Cytometry

BAL and peripheral blood samples will be prepared for analysis using flow cytometry. Samples will be analyzed for T cell, NK cell and neutrophils expression.

## 9.2.3 Gene expression profiling

BAL, and peripheral blood samples will be prepared for the gene array analysis. Specifically, arrays focused on Apoptosis, Dendritic cells/Antigen Presentation, Cytokines,

11-H-0064~Am~L


and Chemokines/Adhesion Molecules will be used. The use of smaller, more focused arrays decreases statistical problems associated with multiple testing and simplifies data analysis. Most interesting and significant findings will be validated by PCR and protein based assays such as immunohistochemistry and ELISA.

- **9.3 Storage:** Research samples will be stored in the secure laboratory of Dr. Richard Childs (NHLBI) and/or Dr. Anthony Suffredini (Clinical Center/Critical Care Medicine Department) under the care and supervision of the principal investigator of this study. All laboratory personnel with access to samples or patient information will complete the NIH online course in Protection of Human Subjects. Efforts to ensure protection of patient information include:
  - The laboratory is located in a controlled access building and laboratory doors are kept locked at all times. Visitors to the laboratory are required to be accompanied by laboratory staff at all times.
  - Hard copy records or electronic copies of documents containing patient information are kept in the locked laboratory or other controlled access locations.
  - An electronic database is used to store information related to patient samples processed by the laboratory.
  - All samples collected will be assigned a unique code.
  - Vials holding patient samples are labeled with the sequential laboratory accession ID number that does not contain any personal identifier information.
  - Samples will be stored until they are no longer of scientific value or until the patient withdraws consent, at which time they will be destroyed.
  - If a patient withdraws consent for their continued use, their sample will be destroyed.
- **9.4 Tracking:** Samples will be ordered and tracked through the CRIS Research Screens. Should a CRIS screen not be available, the NIH form 2803-1 will be completed and will accompany the specimen and be filed in the medical record. Samples will not be sent outside NIH without IRB notification and an executed MTA.
- **9.5** End of study procedures: Samples from consenting subjects will be stored until they are no longer of scientific value or if a subject withdraws consent for their continued use, at which time they will be destroyed. The results will be submitted to the clinicaltrials gov database.
- **9.6** Loss or destruction of samples: Should we become aware that a major breech in our plan for tracking and storage of samples has occurred, the IRB will be notified.

## 10.0 BIOSTATISTICAL CONSIDERATIONS

## 10.1 Primary and secondary endpoints

The *primary objective* is to assess the long-term safety and efficacy of continued therapy with inhaled aerosolized cyclosporine A solution in hematopoietic (group A) and lung transplant patients (group B) with bronchiolitis obliterans (BO) or BO syndrome (BOS) who have shown evidence for a benefit of CIS as previously defined.

Secondary objectives include investigation of the inflammatory pathways that lead to chronic BO and ascertainment of the long term anti-inflammatory effects of this CSA preparation ex vivo and in vivo. Secondary endpoints include improvement of high-resolution CT images, the results of peripheral

11-H-0064 Am L


blood and bronchoalveolar cytokine arrays (secondary markers of inflammation), and the results of functional capacity measurements (pulmonary function tests), and quality of life measurements.

We will evaluate response for group A and group B patients separately, in order to assess if the treatment is effective in each disease.

*Note: As of March 2017 this study is no longer enrolling lung transplant recipients.* 

# 10.2 Sample size

As this is an extension study, the number of patients to be included is directly determined by the number of patients having successfully completed the end of the End of Study (Week 18) visit on companion initial treatment protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans) without evidence of progression of BO. The number cannot exceed 78.

## 10.3 Data Analyses

Any patient who receives any amount of study medication during this extension study will be considered evaluable for safety analysis. Adverse events will be tabulated by severity and disease (lung versus hematopoietic).

Final statistical analysis of efficacy will be performed once all subjects have completed the end of study assessments and all data have been archived for analysis. We will use stratified analyses to account for effects of systemic immunosuppressive agents and other prognostic factors.

## 10.4 Stopping Rule

The study will be monitored to ensure that the occurrence of a specified set of treatment related serious adverse events (TRSAEs) during the subsequent weeks (18-70) of intervention does not substantially exceed an anticipated rate. The following TRSAEs will be considered for early stopping of either one of groups A or B:

- Death considered to be probably or definitely related to the inhaled CsA or
- Any grade IV toxicity considered to be probably or definitely related to inhaled CsA, i.e. opportunistic infection such as tissue-invasive CMV or *Pneumocystis carinii*, with exception of temporary cytopenias.

We will monitor the numbers of subjects who have developed any of the above-specified TRSAEs using the stopping rule outlined below. The trial will be seriously considered for early stopping if the number of subjects in the trial who develop TRSAEs is over the pre-specified threshold value in the Table.

From experience using this agent in other clinical settings as detailed in the investigator's brochure, we anticipate the rate of developing at least one of the above-specified TRSAEs to be 10% or less. Following Geller et al., our stopping rule is determined by a Bayesian approach<sup>23</sup>. The stopping boundary for the trial is reached if the Bayesian posterior probability that the true probability of developing one or more of the above-specified TRSAEs exceeds this benchmark rate of 10% is at least 90%. We take our prior distribution to be a beta distribution with the sum of the two beta

11-H-0064 Am L


parameters to be 3, i.e. the parameters of the beta prior distribution are 0.30 and 2.70. Since we have seen in the past that the first few subjects to be accrued are possibly sicker than the rest of the subjects in the sample, we will start safety monitoring when 3 subjects have developed specified SAEs. The following table summarizes the threshold numbers for stopping either group A or B:

| Number of Subjects | Stop if the number of subjects who develop any of the number of specified TRSAEs reaches: |
|---|---|
| ≤11 | 3 |
| $12 \le n \le 18$ | 4 |
| $19 \le n \le 25$ | 5 |
| $26 \le n \le 32$ | 6 |
| 33 ≤ n ≤ 39 | 7 |

We investigated the performance of the above stopping rules by a simulation study. For the stopping rule, we generated a study with 39 independent Bernoulli trials, each had a probability p=.1 for having the above TRSAE and q=1-p for not having such TRSAE and compared the TRSAE outcomes with the above stopping boundary to determine whether the study was stopped. We repeated the simulation 100,000 times and computed the proportion of stopped studies (i.e. "number of stopped studies"/100,000), which were stopped using the above stopping rule.

The following table summarizes the proportions of stopped studies under a number of scenarios.

| $\boldsymbol{\varepsilon}$ | 1 1 | 11 | | | |
|---|---|---|---|---|---|
| Prob of specified TRSAE | 5% | 10% | 15% | 20% | 30% |
| Proportion of Stopped Studies | 2.2% | 20.2% | 51.5% | 77.4% | 98.1% |
| Average Number of Subjects | 38.4 | 34.5 | 27.8 | 21.0 | 11.9 |
| Average Number of Subjects<br>Suffering TRSAE | 1.93 | 3.47 | 4.18 | 4.18 | 3.54 |

The DSMB will evaluate all serious adverse events and have all the required information to implement the above-defined monitoring plan. In addition, the DSBM may recommend early study termination if other unforeseen adverse events necessitate this decision.

#### 10.5 Off Study Criteria

10.5.1 Patient choice: Subjects may withdraw from the study at their request any time. The risks of withdrawing will be discussed, as will alternative treatment options. Those subjects who choose to withdraw will be strongly encouraged to participate in study assessments until he/she initiates alternative BO therapy. In this scenario, patients will be deemed off study-drug, but have the option to continue on-study.

# 10.5.2 Principal investigator decision:

Subjects will be taken off study drug during study if:

- Subject demonstrates disease progression, as defined by
  - o a 20% or more decline in FEV<sub>1</sub> on two successive measurements at least two weeks apart or

11-H-0064~Am~L


- an increase in the existing dose of one or more immunosuppressive therapies by at least 25% above baseline levels from the primary protocol due to worsening BO/BOS (sustained for 3 weeks, excluding adjustments made for target drug levels) or
- subject requires the addition of new immunosuppressive therapies(sustained for 3 weeks) due to worsening symptoms related to BO/BOS.
- Evidence of an NCI grade IV toxicity related to study drug administration.
- Worsening performance status, defined by ECOG score ≥ 3 (please see hematology supportive care guidelines).
- Disease relapse or a significant non-pulmonary transplant complication in which death is likely to occur and prohibit administration of CIS.
- Patients that have had their CIS tapered off with no worsening of PFTs in the subsequent 12 months.
- Inability to comply with the study visits or become severely ill and cannot comply with the intervention.
- Are unable to tolerate the 150 mg dose of the inhaled CsA.
- Develop severe pulmonary infection that fails to respond to conventional treatment or where no treatment exists.
- Subject becomes pregnant.

These subjects will be asked to complete the end of study assessments, as off-study drug participants, after which they will be referred back to their primary transplant team.

# 10.5.3 Completion of the study

Upon completion of the off study assessments, subjects will have completed study participation and be taken off study and referred back to their primary transplant team to continue post transplant monitoring and care.

## 11.0 DATA AND SAFETY MONITORING PLAN

# 11.1 Safety Monitoring

*Principal Investigator:* Accrual, efficacy and safety data will be monitored by the Principal Investigator, Nicole Gormley, MD and Richard Childs, M.D., Medically Responsible Investigator.

**NIH IntramuralIRB.** Accrual and safety data will be monitored and reviewed annually by the Institutional Review Board (IRB). Prior to implementation of this study, the protocol and the proposed patient consent and assent forms will be reviewed and approved by the properly constituted Institutional Review Board (IRB) operating according to Title 45 CFR 46. This committee will also approve all amendments to the protocol or informed consent, and conduct continuing annual review so long as the protocol is open to accrual or follow up of subjects.

**NHLBI DSMB**: The NHLBI Data Safety and Monitoring Board will review the protocol at an interval to be determined by the DSMB. A progress report will be forwarded to the DSMB at these times and their recommendations will be expeditiously implemented. The DSMB may recommend early termination of the study for considerations of safety and efficacy.

11-H-0064 Am L


**FDA:** An annual progress report, any amendments to the protocol, and any change in the status of the protocol will be forwarded to FDA to:

June Germain, Regulatory Officer
Renata Albrecht, MD, Division Director
Division of Special Pathogen and Transplant Products Central Document Room Center of
Drug Evaluation and Research, FDA
5901-B Ammendale Road Beltsville, MD 20705 (w) 301-796-4024

**APT Pharmaceuticals, Inc.**: An copy of the annual progress report to FDA, any amendments to the protocol, and any change in the status of the protocol will be forwarded to

Greg Baigent [gbaigent@aptbio.com]
APT Pharmaceuticals, Inc
700 Airport Blvd, Suite 350, Burlingame, California 94010
Telephone Number
Fax Number

NIH Radiation Safety Committee (RSC): Because the frequency of CT imaging exceeds that which is standard in this patient population, some of the radiation exposure is therefore determined as indicated for research purposes. The Radiation Safety Form 88-23a which, includes dosimetry calculations for the high resolution CT scans, has been submitted to the Radiation Safety Committee and approved (c/o Sarah Kindrick, M.D., Clinical Protocol Administrator, NIH Radiation Safety Committee 301-496-2253) for initial and triennial RSC review so long as the protocol remains open for patient accrual and intervention.

| | Baseline | On CIS | | | | After wk<br>70 | |
|---|---|---|---|---|---|---|---|
| PROTOCOL TIMEPOINT | Wk 18 | Wk<br>30 | Wk<br>42 | Wk<br>54 | Wk<br>70 | Every 6-12<br>weeks* | End of<br>study |
| High resolution chest CT *if clinically indicated | | | | | | * | |

**Data management:** The PI will be responsible for overseeing entry of data into an in-house password protected electronic system and ensuring data accuracy, consistency and timeliness. The principal investigator, associate investigators, research nurses and/or a contracted data manager will assist with the data management efforts. Data will be abstracted from Clinical Center progress notes as well as from progress notes forwarded from home physicians. Laboratory data from NIH will be imported electronically from CRIS into an in-house clinical trial database. Laboratory values from referring home physicians will be entered into the system.

In order to maintain patient confidentiality, all case report forms, study reports and communications relating to the study will identify patients by assigned patient numbers. Case report forms may serve as source data if needed. All human subjects personally identifiable information (PII) as defined in accordance to the Health Insurance Portability and Accountability, eligibility and consent verification will be recorded. Primary data obtained during the conduct of the protocol will be kept in secure network drives or in approved alternative sites that comply with NIH security standards. Primary and final analyzed data will have identifiers so that research data can be attributed to an individual human subject participant, e.g. a unique code, or minimum PII required for subject identification. All primary and analyzed data will be located on the secure P drive.

11-H-0064 Am L Version Date: 10 May 2019

In accordance with local and federal regulations, the Investigator will allow APT Pharmaceuticals, Inc. personnel or their designee, access to all pertinent medical records in order to verify the data gathered on the case report forms and to audit the data collection process. The US Food and Drug Administration (FDA) may also request access to all study records, including source documentation for inspection.

*End of study procedures*: Data will be stored in locked cabinets and in a password protected database until it is no longer of scientific value. Federal law requires that an Investigator maintain all study records for the indication under investigation for two years following the date a Product Licensing Application is approved or, if no application is to be filed or if the application is not approved for such indication, until two years after the investigation is discontinued and the FDA is notified.

*Clinical Trial Monitoring Plan:* Monitoring Responsible Party/ Monitor: An experienced independent protocol monitoring group has been contracted by the NHLBI. They will objectively audit records for compliance with the protocol.

Monitoring will assure the adequate protection of human subjects, safety of subjects involved in clinical investigations and the integrity and quality of data. The monitor/responsible party for monitoring will be trained to perform monitoring activities.

Monitoring may occur prior to the IRB approval of the study (protocol/ site initiation), routine monitoring (during the protocol life cycle), and study termination. The monitoring activities will verify regulatory compliance, NIH & DIR policy compliance, IRB regulatory compliance, subject record review, and protocol compliance. The monitoring activities will be documented and the reports will be made available to regulatory personnel.

**Loss or destruction of data**: Should we become aware that a major breech in the our plan to protect patient confidentiality and trial data has occurred, the IRB will be notified.

**Publication Policy**: Given the research mandate of the NIH, patient data including the results of testing and responses to treatment will be entered into an NIH-authorized and controlled research database. Any future research use will occur only after appropriate human subject protection institutional approval such as prospective NIH IRB review and approval or an exemption from the NIH Office of Human Subjects Research (OHSR).

#### 12. ADVERSE EVENTS

#### 12.1 Definitions

Adverse Event (AE): Any untoward or unfavorable medical occurrence in a human subject, include any abnormal sign (e.g. abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the research. AE data are recorded on the CRF. The Principal Investigator or a physician member of the research team and the study coordinator will assess each participant for any new or continuing adverse events.

An abnormal laboratory value will be considered an AE if the laboratory abnormality is characterized by any of the following:

• Results in discontinuation from the study

11-H-0064 Am L


- Is associated with clinical signs or symptoms
- Requires treatment or any other therapeutic intervention
- Is associated with death or another serious adverse event, including hospitalization
- Is judged by the Investigator to be of significant clinical impact
- If any abnormal laboratory result is considered clinically significant, the investigator will provide details about the action taken with respect to the test drug and about the patient's outcome.

Serious Adverse Events (SAE): A serious adverse event: Any adverse event that:

- results in death;
- is life-threatening (places the subject at immediate risk of death from the event as it occurred);
- results in inpatient hospitalization or prolongation of existing hospitalization.
- results in persistent or significant incapacity.
- results in a congenital anomaly/birth defect; or based upon appropriate medical judgment, may jeopardize the subject's health and may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.

**Serious event:** An event is serious if it meets the definition of a serious adverse event (above) or if it requires immediate corrective action by a PI and/or IRB to protect the safety, welfare or rights of subjects.

Unanticipated problem that is not an Adverse Event (UPnonAE): An unanticipated problem that does not fit the definition of an adverse event, but which may, in the opinion of the investigator, involves risk to the subject, affect others in the research study, or significantly impact the integrity of research data. For example, report occurrences of breaches of confidentiality, accidental destruction of study records, or unaccounted-for study drug.

**Protocol Deviation (PD):** Any change, divergence, or departure from the IRB approved study procedures in a research protocol that does not have a major impact on the subject's rights, safety or well-being, or the completeness, accuracy and reliability of the study data.

Unanticipated Problem (UP): Any incident, experience, or outcome that is:

- 1. unexpected in terms of nature, severity, or frequency in relation to
  - a. the research risks that are described in the IRB-approved research protocol and informed consent document; Investigator's Brochure or other study documents; and
  - b. the characteristics of the subject population being studied; and
- 2. related or possibly related to participation in the research; and
- 3. places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

#### 12.2 Assessment of Adverse Event Severity and Relationship to Treatment

The AEs will be graded by severity utilizing CTC version 4.0. A copy of the criteria can be downloaded from the CTEP home page at <a href="http://ctep.cancer.gov/reporting/ctc.html">http://ctep.cancer.gov/reporting/ctc.html</a>. The category that overall best "fits" the relationship between the adverse event and the study drug should be chosen and recorded on the CRF and SAE form, if appropriate.

The investigator is responsible for assessing the causal relationship between any events and the study treatment. AEs will be attributed as unrelated, unlikely, possibly, probably, or definitely related to study medication or procedures. Additionally, the investigator is responsible for

 $11\text{-H-}0064\;Am\;L$ 


providing appropriate treatment for the event and for adequately following the event until resolution.

# Relationship Between Treatment and AE

| Unrelated | No temporal association to study product. |
|---|---|
| | An alternate etiology has been established. |
| | The event does not follow the known pattern of response to study |
| | product. |
| | The event does not reappear or worsen with re-challenge. |
| Probably not | No temporal association to study product. |
| related / remote | Event could readily be produced by clinical state, environmental or |
| | other interventions. |
| | The event does not follow the known pattern of response to study |
| | product. |
| | The event does not reappear or worsen with re-challenge. |
| Possibly related | Reasonable temporal relationship to study product. |
| | The event is not readily produced by clinical state, environmental, or |
| | other interventions. |
| | The event follows a known pattern of response to the study product |
| | <u>or</u> as yet unknown pattern of response. |
| Probably related | There is a reasonable temporal association with the study product. |
| | The event is not readily produced by clinical state, environmental, or |
| | other interventions. |
| | The event follows a known pattern of response to the study product. |
| | The event decreases with de-challenge. |
| Definitely related | There is a reasonable temporal relationship to the study product. |
| | The event is not readily produced by clinical state, environmental, or |
| | other interventions. |
| | The event follows a known pattern of response to the study product. |
| | The event decreases with de-challenge and recurs with re-challenge. |

# 12.3 Guidelines Event Reporting

## **Safety Monitoring/Recording/Reporting of Events:**

## **Serious Events**

# Reports to the IRB and CD:

The PI must report serious UPs, and serious PDs, to the IRB and CD as soon as possible but not more than 7 days after the PI first learns of the event.

# Reports to the IRB Chair and CD:

The PI must report all SAEs that do not meet the definition of UP to the IRB chair and CD not more than 14 days after the PI first learns of the event.

# **Non-serious Events**

# Reports to the IRB and CD:

The PI must report all UPs that are not serious to the IRB and CD, and PDs that are not serious to the IRB, not more than 14 days after the PI first learns of the event.

11-H-0064 Am L


#### **Deaths**

The PI must report all deaths (that are not UPs) to the CD as soon as possible, but not more than 7 days after the PI first learns of the event.

#### Reports at the time of continuing IRB review:

At continuing review, the PI will provide to the IRB a summary of:

- All UPs
- All PDs (except for those granted a waiver of reporting)
- All AEs (except for those granted a waiver of reporting)

Clinical adverse events determined directly attributable to the transplant, drugs used in the post-transplant setting, and progression of baseline disease for which the transplant was indicated will not be collected; however these events will be recorded in the patient's medical record.

Adverse laboratory events used to evaluate the safety of this protocol regimen will be collected to include any change from laboratory assessments done prior to first dose of study medication that result in a progression to a grade 3 or 4 laboratory toxicity.

Abnormal labs determined directly attributable to the transplant, drugs used in the post-transplant setting, and/or progression of baseline disease for which the transplant was indicated will not be collected; however these events will be recorded in the patient's medical record.

Only serious and unexpected adverse events related to this protocol will be reported on this ancillary study. Those determined serious and unexpected adverse events related to post transplant complications will be reported on the transplant protocol.

**Treatment related SAEs (TRSAEs)** are those attributed as possibly, probably or definitely. As detailed in section 10.4 stopping rules, death and any grade IV toxicity considered to be possibly, probably or definitely related to inhaled CIS will be monitored and considered for early stopping the study according to statistically determined criteria.

Hospitalization (overnight admission) for routine supportive care (platelet or RBC transfusions) or admission from the NIH inpatient unit to the NIH ICU for routine monitoring will not be reported as a serious adverse event.

Unanticipated problems that are either AEs or non-AEs, (as defined by Section 12.1 above) will be reported within 7 calendar days of investigator awareness.

All serious adverse events will also be distributed to the Data Safety Monitoring Committee within the same timeframe required for IRB reporting of SAEs.

**APT Pharmaceuticals, Inc.**: A listing of all SAEs will be submitted to APT pharmaceutical quarterly. Safety reports will be reported as detailed in section 12.5.

## 12.4 IND Safety Reporting to the FDA (IND 109,707)

Because this study will be conducted under an IND, U.S. Government regulations 21CFR, Part 312.32 require the issuance of an IND Safety Report to the Food and Drug Administration (FDA) for all "serious" adverse events that are "unexpected" and for which there is a "reasonable

 $11\text{-H-}0064\;Am\;L$ 


possibility that the experience may have been caused by the drug." Such serious events that are characterized as fatal or life-threatening must be reported to the FDA within 7 calendar days of the sponsor's initial receipt of the information, whereas non-fatal and non-life threatening events must be reported within 7 calendar days.

No expedited IND Safety Report is required if the event is considered to be expected based either on the study drug product label, the underlying disease states, or the study procedures.

The Safety report will contain a full written summary detailing relevant aspects of the serious adverse events in question. In each written IND safety report, all safety reports previously filed with the IND concerning a similar adverse experience will be included and the significance of the adverse experience in light of the previous, similar reports will be discussed.

Where applicable, information from relevant hospital case records and autopsy reports will be included. The investigator will always provide an assessment of causality at the time of the initial report as described in 'Assessment of Causality'.

Follow up information regarding the patient's subsequent course will be submitted until the SAE has resolved, the patient's condition stabilizes (in the case of persistent impairment) or the patient dies.

Reports from animal studies will be submitted in a narrative format.

# 12.5 Sponsor's Reporting Responsibilities

Serious and unexpected suspected adverse reactions (SUSARs) as defined in 21 CFR 312.32 and determined by the sponsor will be reported to FDA as IND Safety Reports. The Sponsor will also submit an IND Annual Report of the progress of the investigation to the FDA as defined in 21 CFR 312.33.

Telephone and facsimile transmission safety reports. The sponsor shall also notify IRB, DSMB APT and FDA by telephone or by facsimile transmission of any **unexpected fatal or life-threatening experience associated with the use of the drug** as soon as possible but in no event later than 7 calendar days after our initial receipt of the information.

Hard copy submission of safety reports: Each notification will be made as soon as possible and in no event later than 7 calendar days after the sponsor's initial receipt of the information.

If an adverse drug experience not initially determined to be reportable is later determined reportable, a written safety report will be submitted as soon as possible, but in no event later than 7 calendar days after the determination is made.

# 12.5.1 Report Recipients

Safety reports will be submitted according to the reporting time frame (section 21.5) to

- NHLBI IRB
- NHLBI DSMB

 $11\text{-H-}0064~\mathrm{Am}~\mathrm{L}$ 


- FDA: June Germain, Regulatory Officer
   Renata Albrecht, MD, Division Director
   Division of Special Pathogen and Transplant Products Central Document Room
   Center of Drug Evaluation and Research, FDA
   5901-B Ammendale Road, Beltsville, MD 20705 (w) 301-796-4024
- APT APT pharmacovigilance Officer APT Pharmaceuticals, Inc 700 Airport Blvd, Suite 350, Burlingame, California 94010

## 12.6 Reporting of pregnancy

Subjects who become pregnant during the study will discontinue the study medication immediately. The investigator, or his/her designee, will collect pregnancy information on any subject who becomes pregnant while participating in this study and submit this information to APT and the IRB within two weeks of learning of a subject's pregnancy. Information on the status of the mother and fetus will be forwarded to APT and the IRB as available. While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication, spontaneous abortion, or elective termination of a pregnancy for medical reasons will be reported to APT in an SAE format. Generally, follow-up will be no longer than 6 to 8 weeks following the estimated delivery date and will include information on outcome of the pregnancy.

# 13.0 HUMAN SUBJECT PROTECTIONS

# 13.1 Rationale for Subject Selection

Subjects will be considered eligible if they have completed the 19-week assessment on the initial protocol (Phase II Trial of CIS in lung transplant and hematopoietic stem cell transplant recipients for treatment of Bronchiolitis Obliterans) and show either an improvement or stabilization in BO/BOS with CIS treatment defined by the above inclusion/exclusion criteria.

From previous hematopoietic transplant protocol recruitment patterns from NHLBI transplant recipients, we expect the population accrued from the companion initial treatment protocol may be distributed as follows:

- By gender: 40% females; 60% males
- By age: ages 11-73, median 38; 7% ages 10-17; 20% ages 18-30; 28% ages 31-40; 22% ages 41-50 and 23% ages 51-73
- By race: 11% Asian, 8% Black, 44% Hispanic, 37% White

The Lung transplant recipients participating on the companion initial treatment protocol may be distributed as follows:

By gender: 45% females; 55% males
By age: ages 23-71, median 58
By race: 45% Black, 55% White

**Recruitment:** Subjects will be recruited from those subjects who have completed participation on companion initial treatment protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in

11-H-0064 Am L


Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans) and meet long-term study inclusion/exclusion criteria.

Competition with other Branch protocols: None. However, there is an actively accruing protocol at the Clinical Center 08-C-0097: A Multi-Institutional Prospective Phase II Study of Montelukast for the Treatment of Bronchiolitis Obliterans Following Allogeneic Stem Cell Transplantation in Children and Adults. They will refer patients to our study that have completed/failed their protocol.

**Reimbursement for protocol participation, travel, food, and lodging** will be consistent with NIH guidelines. In determining reimbursement, the following factors are considered applicable to this protocol: the patients are diagnosed with a rare disease; the patient population is sick; the protocol offers the potential for direct benefit; the protocol regimen is demanding; and in order to complete accrual in a reasonable timeframe a geographically dispersed participant population is required.

Note: As of March 2017 this study is no longer enrolling lung transplant recipients.

## 13.2 Participation of Children

This study will be limited to subjects aged 10 or older. Various study tests and medication administration requires adequate understanding and ability to participate in care. As such, pediatric patients 10 years of age or older will be allowed to participate in this study as they are at an age where they can cooperate sufficiently and children less than age 10 will be excluded.

#### 13.3 Risks and Discomforts

#### 13.3.1 Related to Inhaled CIS

CIS is under development for the indication of improved BOS-free survival following lung transplantation. As of November 13, 2009, approximately 444 lung transplant recipients have received CIS under protocols ACS001, ACS002, ACS004, or CIS001. n ACS001, the following adverse events occurred significantly more often in patients receiving CIS than in patients receiving placebo:

- Events that occurred in 30 to 50% of patients receiving CIS: cough, chest pain, back pain, increased urinary frequency, pharyngitis, exacerbation of shortness of breath, and lung consolidation.
- Events that occurred in 10 to 29 % of patients receiving CIS: cardiac murmur, respiratory tract irritation, polyuria, somnolence, hyperlipidemia, respiratory disorder, and hemoptysis.

In the studies that were not placebo controlled, or are as yet unblinded, the following adverse events were seen:

• Events that occurred in greater than 10% of patients: pyrexia, nausea, diarrhea, dyspnea, cough, wheezing, chest pain, pharyngitis, renal impairment, peripheral edema, lung transplant rejection, headache, insomnia, and neutropenia.

 $11\text{-H-}0064\;Am\;L$ 


• Events that occurred in 5 to 10% of patients: Pharyngolaryngeal pain, pleural effusion, rhinorrhea, constipation, vomiting, fatigue, chest pain, candidiasis, pseudomonas infection, sinusitis, pneumonia, hyperkalemia, leucopenia, anemia, and hypertension.

Although not previously observed, in the initial phase of the NIH study, one subject did develop a rib fracture associated with coughing.

Unknown side effects: In addition, as with other clinical studies using experimental medicines and in subjects with serious medical conditions, there may be adverse events or side effects that are currently unknown and certain of these unknown risks could be permanent, severe, or life threatening. Subjects will therefore be carefully monitored and instructed to seek medical attention in the event of serve adverse events and contact the research team as needed.

Cyclosporine, when taken by mouth can cause kidney damage especially if blood levels are high. So far, use of CIS has not caused this problem in previous human research studies and should not increase this risk since blood levels have been very low.

APT Pharmaceuticals remains attentive to safety throughout all ongoing studies. Additional unexpected safety findings will be provided to investigators upon receipt and evaluation.

#### 13.3.2 Related to albuterol/levalbuterol

Severe allergic reactions (rash; hives; itching; difficulty breathing; tightness in the chest; swelling of the mouth, face, lips, or tongue); chest pain; ear pain; fast or irregular heartbeat; new or worsened trouble breathing; pounding in the chest; red, swollen, blistered, or peeling skin; severe headache or dizziness; unusual hoarseness; wheezing. Subjects will be instructed to discontinue albuterol/levalbuterol use, seek medical attention right away, and notify the research teams should any severe side effect occur.

The most common side effects include: Dizziness; headache; nausea; nervousness; sinus inflammation; sore or dry throat; tremor; trouble sleeping; vomiting.

#### 13.3.3 Related to blood collection

Blood collection my cause some pain or bruising at the site on the arm from which the blood was drawn. There is a small possibility of fainting and infection. Similarly, there is a small risk of bleeding, blockage, or inflammation or infection of the vessel. Discomfort does not usually last long and permanent damage is extremely rare.

## 13.3.4 Related to Bronchoalveolar Lavage (BAL)

Subjects will sign a separate procedure consent for the BAL which will further detail the potential risks of this procedure which include:

- Mild discomfort due to coughing. This can be controlled by topical medication.
- A decrease in the amount of oxygen in the blood. Subjects will receive additional oxygen during the procedure and they will be closely monitored for oxygen levels, heart rate and blood pressure. The risk of a serious problem occurring is very small (less than 1 out of 10,000 procedures in published studies).

 $11\text{-H-}0064\;Am\;L$ 

- A slow or irregular heartbeat occurs (rare). If it does not correct itself, we can treat this with medication. A heart rhythm monitor (electrocardiograph) will be used throughout the procedure.
- Mild bleeding from the nose can occur because the bronchoscope tube is sometimes placed through the nose to reach the large airways. Placing medication and lubricant inside the nose will be done before the procedure to lower the risk of this occurring.
- A sore throat for several hours after the procedure (less than 10% of patients).
- A bad reaction to the numbing medication (lidocaine), rarely. Side effects can include confusion or, very rarely, seizures. We have never seen this problem in over 1500 bronchoscopies performed in the Medical Intensive Care Unit at NIH over an 8-year period. This potential problem is minimized by using small, frequent doses of the medication.
- Fever has been reported to develop in less than 5% of healthy volunteers six to eight hours after the bronchoscopy.
- Infection in the lungs (very low risk) resulting from swallowing saliva into the lung airways. To minimize this risk, subjects do not eat or drink for at least six hours before the bronchoscopy.
- Individuals with lung disease may be at greater risk of complications from bronchoscopy, although bronchoscopies with bronchoalveolar lavage are performed commonly for such patients without any serious complications or effects.
- There are risks associated with the conscious sedation medicine. These risks will be explained to the subjects and they will be consented separately at the time of the procedure.

#### 13.3.5 Related to the Lung Function Tests:

These tests are very safe and side effects are unlikely. During the test, subjects are asked to breathe deeply or rapidly, which may occasionally cause brief lightheadedness or soreness of the chest. In extremely rare cases, this may result in the release of a small amount of air from the lung into the lung cavity, which would be treated appropriately.

#### 13.3.6 Related to the 6 Minute Walk

Subjects may develop shortness of breath or fatigue. Participants will be encouraged to walk at a pace that is comfortable for them.

#### 13.3.7 Related to Pregnancy and Nursing Mothers

The effects of albuterol and/or aerosolized cyclosporine A in solution with propylene glycol on the developing human fetus are unknown. For this reason and because it is unknown whether these drugs are teratogenic, women of childbearing potential and men must agree to use adequate contraception prior to (hormonal or barrier method of birth control; abstinence) and for the duration of study participation. If a woman becomes pregnant or suspects she is pregnant while on study,

 $11\text{-H-}0064\;Am\;L$ 


her treating physician should be informed immediately. Nursing mothers must be willing to discontinue nursing.

### 13.3.8 Related to the high resolution CT (radiation):

CT (computed tomography), sometimes called CAT scan, uses special x-ray equipment to obtain image data from different angles around the body and then uses computer processing of the information to show a cross-section of body tissues and organs. Oral and/or intravenous contrast agents will NOT be used.

#### 13.4 Risks in relation to benefits

#### 13.4.1 For Adult Subjects

The risks of participating in this trial are limited to side effects of the albuterol/levalbuterol and inhaled CsA, and the risks of standard diagnostic procedures (BAL and biopsy, the high resolution CT, and pulmonary function tests), the 6 minute walk, and the additional peripheral blood sample to be used strictly for research purposes. Samples for clinical monitoring will be collected during sample collection procedures that are part of their routine post transplant care and therefore pose no additional burden or risk.

The benefits to the subjects could be improvement in BO resulting in improved quality of life, decreased mortality associated with severe BO (should it develop), and potentially, treatment with other more toxic systemic therapies could also be avoided or postponed. Subjects will also receive direct health benefits due to thorough post transplant pulmonary examinations, early diagnosis of progression of BO and therefore earlier access to appropriate BO management. Therefore, for adult subjects participating on this study, the research involves greater than minimal risk to subjects with the prospect of direct benefit (45 CFR 46.102).

As of May 10, 2019, this study is now closed to new subject accrual and continues in data analysis and/or sample analysis only and the level of risk is now minimal.

#### 13.4.2 For pediatric subjects

DHHS will conduct or fund research in which the IRB finds that more than minimal risk to children is presented by an intervention or procedure that holds out the prospect of direct benefit for the individual subject, only if the IRB finds that:

- (a) "The risk represents a minor increase over minimal risk". The risks of participating in this trial are limited to the side effects of the albuterol and inhaled CsA, the risks of standard diagnostic procedures (BAL and biopsy, the high resolution CT, the pulmonary function tests and the 6 minute walk), and the additional peripheral blood sample to be used strictly for research purposes. Samples for clinical monitoring will be collected concurrently with samples that are part of their routine post transplant care. Only those laboratory tests approved by the IRB and involving not greater than minimal risk will be conducted (See Appendix B).
- (b) The relation of the anticipated benefit to the risk is at least as favorable to the subjects as that presented by available alternative approaches. The risk associated with the monitoring that will be done on this ancillary protocol exceeds only minimally that would be done routinely in post transplant patients who have developed BO. This risk is most favorable given that pediatric subjects could derive benefit in improvement in BO, resulting in improved quality of life,

 $11\text{-H-}0064\;Am\;L$ 


decreased mortality associated with severe BO (should it develop), and avoidance of treatment with other more toxic systemic therapies. Subjects will also receive direct health benefits due to thorough post transplant pulmonary examinations, early diagnosis of BO progression, and therefore earlier access to appropriate BO management.

(c) Adequate provisions are made for soliciting the assent of the children and permission of their parents or guardians, as set forth in 46.408. An assent is available.

Therefore, the inclusion of children satisfies the criteria set forth in 45 Code of Federal Regulations 46, Subpart D: 46.405 Research involving greater than minimal risk but presenting the prospect of direct benefit to the individual subjects.

#### 13.5 Informed Consent Processes and Procedures

The investigational nature and research objectives of this trial, the procedure and its attendant risks and discomforts will be carefully explained to the subject and when applicable the subjects' parents. The potential subject will be educated regarding the nature of the condition, proposed intervention, and outcome measures. Study subjects will be informed that participation is entirely voluntary and that withdrawal from the study can be made at any time without penalty of benefits to which they may be entitled. No consenting will be done by outside investigators or at outside institutions.

At any time during participation in the protocol, if new information becomes available relating to risks, adverse events, or toxicities, this information will be provided orally or in writing to all enrolled or prospective patient participants. Documentation will be provided to the IRB and if necessary the informed consent amended to reflect relevant information.

**Informed consent of non-English speaking research participants:** We anticipate the enrollment of Spanish-speaking research participants into our study. The IRB approved full consent document will be translated into that language in accordance with the Clinical MAS Policy M77-2. If there is an unexpected enrollment of a research participant for which there is no translated extant IRB approved consent document, the principal investigator and or those authorized to obtain informed consent will use the Short Form Oral Consent Process as described in MAS Policy M77-2, 45 CFR 46.117 (b) (2), and 21 CFR50.27 (b) (a). The summary that will be used is the English version of the extant IRB approved consent document.

We request prospective IRB approval of the use of the short form for up to a minimum of 10 participants in a given language and will notify the IRB at the time of continuing review of the frequency of the use of the Short Form. Should we reach the threshold of 10, we will notify the IRB of the need for an additional use of the Short Form and that we will have that consent document translated into the given inherent language.

Minor patients: If the patient is a minor, a minor assent will be sought. Where deemed appropriate by the clinician, and the child's parent or guardian, the child will also be included in all discussions about the trial and a minor's assent will be obtained. The parent who signs the consent for the minor must be a legally recognized parent or guardian. The parent or guardian will sign on the designated line on the informed consent attesting to the fact that the child had given assent. When the assent is not age appropriate, the study will be explained to the child and the assent will

11-H-0064 Am L Version Date: 10 May 2019

be obtained verbally from the child. Once the minor reaches 18, he/she will be consented for continued protocol participation using the adult consent.

Because this research holds a prospect of direct benefit to the health or well-being of pediatric participants and is available only in the context of the research, the assent of the pediatric participant is not a necessary condition for proceeding with the research. However, in the case of dissent, an independent pediatric care team (social worker and mental health specialist (psychologist or psychiatrist) will meet with the minor and his family to re-emphasize the importance of treatment on protocol; if the child continues to dissent, an ethics consult will be requested prior to enrollment.

When a pediatric subject reaches age 18, continued participation will require re-consenting of the now adult with the standard protocol consent document to ensure legally effective informed consent has been obtained. Should sample or data analysis continue following completion of active participation and the subject has reached 18 years of age, we will attempt to contact the subject using the last known contact information to obtain consent for continued use of data or samples collected during their prior visit. Given the length of time that may have transpired for some of the subjects since their last visit for this study, we request waiver of informed consent for those individuals who after good faith efforts to contact them, we are unable to contact.

Requirements for Waiver of Consent consistent with 45 CFR 46.116 (d), each of which must be addressed in relation to the protocol:

- (1) The research involves no more than minimal risk to the subjects;
  - a) Analysis of samples and data from this study involves no additional risks to subjects.
- (2) The waiver or alteration will not adversely affect the rights and welfare of the subjects;
  - a) Samples and data will be kept in secure locations in the laboratory of Dr. Young. Retention of samples or data does not affect the welfare of subjects.
- (3) The research could not practicably be carried out without the waiver or alteration; and
  - a) Considering the length of time between a minor's enrollment and their age of majority, it is possible that more than a few subjects may be lost to follow up. A significant reduction in the number of samples analyzed could impact the quality of the research.
- (4) Whenever appropriate, the subjects will be provided with additional pertinent information after participation.
  - a) We only plan to request a waiver of re-consent for those subjects who have been lost to follow-up.

In cases where parents share joint legal custody in making medical decisions of their child (e.g. by a custody agreement or court order) both parents must give their parental permissions regardless of level of risk of the research. Exceptions may be made if one parent is deceased, becomes incompetent or is not reasonably available (e.g. in prison).

Consenting to Pregnancy Testing in Minors of Childbearing Age: We will inform the minor during the assent process that for safety, we need to do a pregnancy test. She will also be told that if it is positive, we will counsel her and help her tell her parents. If the minor does not want to proceed she will be advised not to sign the assent and her enrollment on this screening protocol will end.

#### 13.6 Conflict of Interest

11-H-0064 Am L


The Principal Investigator assured that each associate investigator listed on the protocol title page received a copy of the NIH's Guide to preventing conflict of interest. Investigators added subsequent to the initial circulation were provided a copy of the document when they were added. No initial or subsequent members of the research team reported a potential conflict of interest.

This protocol has no associated patents, however, outside associate investigator Aldo Iacono, MD holds a US patient application A32130-072396.0162 (11/11/1999) for "Uses of Aerosol Cyclosporine for Prevention and Treatment of Pulmonary Disease". Dr. Timothy Corcoran has received research grant funding from APT through the University of Pittsburg. To avoid any conflict of interest, Drs. Iacono and Corcoran will not participate in the consent process nor will they participate in any of the endpoint evaluations.

### 13.7 Technical Transfer Agreements

This protocol has no associated patents

An MTA with APT Pharamceuticals, Inc was previously signed that allowed for in vitro assays to be performed using the cyclosporine in propylene glycol.

A CRADA between APT Pharmaceuticals, Inc has been fully executed.

#### 14.0 PHARMACEUTICAL

#### 14.1Cyclosporine Inhalation Solution (CIS)

**Physical, chemical, and pharmaceutical properties:** CIS is a sterile, clear, colorless, preservative-free solution of cyclosporine (USP) in propylene glycol developed specifically for administration by oral inhalation. The active principle of CIS is a cyclic polypeptide immunosuppressant agent consisting of 11 amino acids. It is produced as a metabolite by the fungus species Beauveria nivea. The molecular formula is  $C_{62}H_{111}N_{11}O_{12}$  and the molecular weight is 1202.63.

*Chemical name:* The chemical name for cyclosporine is  $[R-[R^*,R^*-(E)]]$ -cyclic(L-alanyl-D-alanyl-N-methyl-L-leucyl-N-methyl-L-valyl-3-hydroxy-N,4-dimethyl-L-2-amino-6-octenoyl-L- $\alpha$ -amino-butyryl-N-methylglycyl-N-methyl-L-leucyl-L-valyl-N-methyl-L-leucyl).

Chemical Structure

11-H-0064 Am L


Supply: CIS is manufactured and filled into a sterile, single-use clear 6 mL glass vial sealed with a sterilized, siliconized light gray bromobutyl rubber stopper secured by a crimped tear-off aluminum overseal. This container closure system provides protection of the formulation from microbial contamination, moisture ingress, and other environmental contaminants during storage. Each vial contains 5.2 mL of solution containing 325 mg cyclosporine. This vial contains a sufficient amount of cyclosporine, USP in propylene glycol, USP to deliver 300 mg in 4.8 mL. CIS is designed specifically for aerosol inhalation via a single use SideStream<sup>®</sup> disposable nebulizer (Respironics, Inc., Murrysville, PA) with the Mobilaire compressor (Invacare, Elyria, OH) at 30 psi. Previous studies have used the AeroTech™ II nebulizer with a high flow compressor such as the Sunrise DeVilbiss 8650D set at 40 pounds per square inch (PSI). At 40 PSI, the average flow rate from the compressors is approximately 12.5 L/min.

**Storage**: CIS vials should be stored in the upright position at controlled room temperature at controlled room temperature, 25°C (77°F), excursions permitted to 15°-30°C (59-86°F). Do not store in the refrigerator or freezer. CIS vials are single use. Any remaining CIS in the vial after dosing should be discarded.

#### **Drug Product Composition**

| Component | Quality<br>Standard | Function | Amount per vial | Concentration<br>(% w/vol) |
|---|---|---|---|---|
| Cyclosporine | USP | Active ingredient | 325 mg | 62.5% |
| Propylene Glycol | USP | Solvent | 5.2 mL | - |

At a formulation of 62.5 mg/mL, the cyclosporine concentration in CIS is well below the saturation solubility of 400 mg/mL in propylene glycol. Cyclosporine is freely soluble at the manufacturing conditions of 20 - 40°C and during long-term storage at 30°C. Therefore, the risk of crystallization during its shelf-life is low.

 $11\text{-H-}0064\;Am\;L$ 


Aerosol Properties: An in vitro study was performed to assess the aerosol characteristics of CIS in the Sidestream® Disposable nebulizer. The mass median aerodynamic diameter (MMAD) particle size was determined by NGI impaction to be 1.9  $\mu$ m. The geometric standard deviation (GSD) was 1.9. These aerosol particle properties are well suited for both large airway and small airway deposition.

**Shipping:** The NIH Pharmaceutical Development Services will be responsible for receiving, storing, dispensing and accounting for drug product. The shipping address for APT Pharmaceuticals, Inc supplied investigational agent is:

National Institutes of Health
PHARM DEV SVC, Room 1D35
10 Center Drive, MSC 1196, Building 10
Bethesda, Maryland 20892-1196
Shipping Designee Name: Judith Starling, RPh

Shipping Designee Phone No: (301) 496-1031 Shipping Designee FAX No: (301) 402-3268 Shipping Designee e-mail: jstarling@NIH.gov

Accountability Procedures: Drug accountability records will be maintained for all clinical supplies. All empty and partially used vials and clinical trial supplies will be destroyed locally according to the institution's standard operating procedures for drug destruction. The pharmacy will maintain detailed documentation of the number and identification of vials, which are destroyed, and copies of these documents will be provided to the Sponsor. Disposition of all unused boxes of study drug will be carried out according to instructions provided by the Sponsor at the end of the study after drug accountability is performed by the study monitor.

#### 14.2 Albuterol

**Physical, chemical, and pharmaceutical properties:** Albuterol is a white or practically white powder, freely soluble in water and slightly soluble in alcohol. It is a relatively selective beta-2 adrenergic bronchodilator. The molecular formula is  $(C_{13}H_{21}NO_3)_2 \cdot H_2SO_4$  and the molecular weight is 576.71.

*Chemical name:* The chemical name for albuterol is  $\alpha^1[(tert\text{-Butylamino})\text{methyl}]\text{-4-hydroxy-m-xylene-}\alpha, \alpha' diol sulfate (2:1) (salt).$ 

#### Chemical Structure:

*Supply:* Albuterol is supplied in unit-dose vials containing albuterol sulfate inhalation solution 0.083%, 2.5mg/3ml.

**Storage**: Albuterol should be protected from light and stored in the pouch until time of use. It should be stored between 2° and 25° C (36° and 77° F).

11-H-0064 Am L


#### 15.0 **ROLE OF COLLABOATORS**

Aldo T. Iacono, M.D., Medical Director, Lung Transplant Program

Role: Will provide advice regarding administration of the CIS, trial design and clinical management of patients who have received a lung transplant

Michael Terrin, MD, Professor of Epidemiology and Medicine

Role: Will provide trial design advice

Timothy Corcoran, PhD, Professor of Medicine and Bioengineering, Pulmonary, Allergy and Critical Care Medicine,

Role: Will provide advice regarding the lung deposition studies

11-H-0064 Am L

PI: N. Gormley


#### 16.0 REFERENCES

- 1. Trulock EP, Edwards LB, Talyor DO, et al. Registry of the International Society for Heart and Lung Transplantation: Twenty-third official adult lung and heart-lung transplantation report-2006. Journal of heart and lung transplantation 2006, 25:880-92
- 2. Savani, BN et al. Chronic GVHD and pretransplantation abnormalities in pulmonary function are the main determinants predicting worsening pulmonary function in long-term survivors after stem cell transplantation. Biology of Blood and marrow transplantation 2006, 12(12):1261-9.
- 3. Afessa B, Litzow M, Tefferi A. Bronchiolitis Obliterans and other late onset pulmonary complications in hematopoietic stem cell transplantation. Bone Marrow Transplantation 2001, 28:425-34
- 4. Bryant D, Obliterative bronchiolitis in haematopoietic stem cell transplantation:can it be treated? European Respiratory Journal 2005, 25:402-04
- 5. Watkins T, Chien J, Crawford S. Graft versus host associated pulmonary disease and other idiopathic pulmonary complications after hematopoietic stem cell transplant. Seminars in respiratory and critical care medicine 2005, 26(5):482-89
- 6. Estenne M, Hertz M. Bronchiolitis Obliterans after human lung transplantation. American journal of respiratory and critical care medicine 2002, 166: 440-44
- 7. Filipovich et al. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. Diagnosis and Staging Working Group Report. Biology of Blood and Marrow Transplantation 2005; 11:945-955
- 8. Iacono AT, Johnson BA, Grgurich WF, et al. A randomized trial of inhaled cyclosporine inlung-transplant recipients. New England journal of medicine 2006, 354(2):141-50
- 9. Boehler A, Estenne M. Post-transplant bronchiolitis obliterans. European respiratory journal 2003, 22:1007-1018.
- 10. Soubani AO, Uberti JP. Bronchiolitis obliterans following haematopoietic stem cell transplantation. European respiratory journal 2007, 29:1007-1019
- 11. Sanchez et al. Long-term follow-up of immunosuppressive treatment for obstructive airways disease after allogeneic bone marrow transplantation. Bone Marrow Transplantation 1997; 20: 403-8
- 12. Burckart et al. Journal of clinical Pharmacology 1989; 29:860
- 13. Mitruka et al. Journal of Thoracic and Cardiovascular Surgery 1998;115(1): 28-36
- 14. Dowling et al. Surgery 1990;108(2): 198-204
- 15. Iacono et al. Aerosolized cyclosporine in lung recipients with refractory chronic rejection. American Journal of Respiratory and Critical Care medicine 1996;153 (4):1451-5

 $11\text{-H-}0064\;Am\;L$ 


- 16. Iacono et al. Aerosol cyclosporin therapy in lung transplant recipients with bronchiolitis obliterans. European Respiratory Journal 2004;23:384-90
- 17. Iacono et al. Transplantation 1997;64:263
- 18. Iacono et al. Dose-related reversal of acute lung rejection by aerosolized cyclosporine. American Journal of Repiratory and Critical Care medicine 1997;155 (5):1690-8
- 19. Keenan et al. Treatment of refractory acute allograft rejection with aerosolized cyclosporine in lung transplant recipients. Journal of Thoracic and Cardiovascular Surgery 1997;113(2):335-40
- 20 Simon R. Optimal two-stge designs for phase II clinical trials. Controlled Clinical Trials 10:1-10, 1989.
- 21. Anhøj et al. Lung deposition of inhaled drugs increases with age. American Journal of Respiratory and Critical Care Medicine 2000;162:1819-22
- 22. Burckart et al. Lung deposition and pharmacokinetics of cyclosporine after aerosolization in lung transplant patients. Pharmaceutical Research 2004: 20(2):252-56
- 23. Geller NL, Leifer ES, Follmann D. and Carter SL. Design of Early Trials in Stem Cell Transplantation: A Hybrid Frequentist-Bayesian Approach. *Advances in Clinical Trial Biostatistics*. 2004.
- 24. Rosenfeld S, Follman D. Nunez O, Young NS. Antithymocyte globulin and cyclosporine for severe aplastic anemia: associated between hematologic response and long-term outcome. JAMA. 2003 Mar 5:289 (9):1130-5)


## **APPENDIX A** MEDWATCH Form FDA 3500A

 $\underline{http://www.fda.gov/Safety/MedWatch/HowToReport/DownloadForms/default.htm}$ 

11-H-0064 Am L Version Date: 10 May 2019

# APPENDIX B NHLBI HEMATOLOGY BRANCH LABORATORY RESEARCH STUDIES v 2/5/2013

| | DESCRIPTION OF LABORATORY STUDY BY BRANCH SECTION | Does this test<br>pose a greater<br>than minimal<br>risk to<br>pediatric<br>subjects per 45<br>CFR 46.404? | pose a greater<br>than minimal<br>risk to<br>healthy<br>pediatric |
|---|---|---|---|
| A | Stem Cell Allotransplantation Section (Dr. A. John Barrett) | | |
| A.1 | Measurement of lymphocyte function and immune responses directed toward allogeneic tissues, malignant cells, and infectious agents. Assay of a variety of antigens, including standard proliferation, cytotoxicity, and intracellular cytokine detection including GVHD predictive markers. Measurement of antigen-specific responses including employment of tetramers, ELISPOT technique, gene amplification-based assays, and flow cytometry. Selection of cells using immunomagnetic beads or flow cytometry. Culture, expansion, and selection of cells. Surface marker analysis of PB MC using flow cytometry. Cytokine/chemokine analysis of plasma/serum samples using ELISA and/or Luminex techniques. | No | No |
| A.2 | Generation of cell lines for the study of immune cell interactions with other cells. Transformation of B-lymphocytes using Epstein-Barr virus. Derivation of malignant cell lines from patient leukemic or solid tumor samples. | No | No |
| A.3 | Infection of cells and cell lines with recombinant genes to ascertain the effects of expressed molecules on immune responses and on growth and development. Transfection of cell lines with specific molecules to study antigen-specific responses. | No | No |
| A.4 | Assays of peripheral blood and bone marrow progenitor cells including primitive and late erythroid progenitor-derived colonies, myelomonocytic colonies, and primitive multi- potential progenitor-derived colonies. | No | No |
| A.5 | Injection of human cells into experimental animals to study the immune system and the growth of normal and malignant cells under varying conditions. | No | No |
| A.6 | Testing of selection methods, cell isolation, and cell expansion leading to the development of new cell-based therapies requiring scale-up for clinical application. | No | No |
| A.7 | Identification of individual T cell clones by their T cell receptor sequence. | No | No |
| A.8 | Measurement of tumor and tissue specific antigens in cells of subjects and donors by mRNA,protein, or peptide expression in cells or fluids. | No | No |
| A.9 | Laser capture micro dissection of cells from biopsies for GVHD to determine clonotypes. | No | No |
| A.10 | DNA and RNA typing of genes that control immune responses in lymphocytes. | No | No |
| A.11 | Microassay studies utilizing cellular DNA, cDNA, and RNA for neoplasia and host-tumor interactions. | No | No |
| В | Molecular Hematopoiesis Section (Dr. Cynthia Dunbar) | | |
| B.1 | Flow cytometric analysis of cell surface and cytoplasmic proteins, including cell adhesion molecules, putative retroviral receptors, and markers of differentiation, using bone marrow and mobilized peripheral blood cells. | No | No |

11-H-0064 Am L


| B.2 | Hematopoietic progenitor-derived colony ascertainment in vitro (as described above), and engraftment of immunodeficient mice for detection of human stem cell number | No | No |
|---|---|---|---|
| B.3 | and function. Testing ability of hematopoietic progenitor cells to be transduced with retroviral, | No | No |
| | lentiviral, and novel gene transfer vectors in vitro. | | |
| B.4 | Reprogramming of adult mature cells, including skin fibroblasts and blood cells, into induced pluripotent stem cells in vitro. | No | No |
| 7 | Call Picture Continue (Do. Mart Versia) | | |
| <u> </u> | Cell Biology Section (Dr. Neal Young) | | |
| C <b>.1</b> | Studies of blood and bone marrow hematopoietic progenitor numbers, including early and late erythroid progenitors, myelomonocytic progenitors, and multi-potential progenitor cells. In addition, bone marrow may be placed in long-term bone marrow culture to assess the function of stroma and stem cells and to assay more primitive progenitors, as well as organelle culture. Whole or selected bone marrow populations are cultured short-term for CD34 cell expansion. | No | No |
| C.2 | Assays of apoptosis in hematopoietic cells and their progeny, using flow cytometric methods such as annexin and caspase-3 staining, propidium iodide uptake, and mitochondrial permeability tests. | No | No |
| C.3 | Separation and functional study of cell populations characteristic of paroxysmal nocturnal hemoglobinuria, identified by absence of glycosylphosphatidylinositol anchored proteins. | No | No |
| C <b>.4</b> | Studies of mutation rates in hematopoietic cells and in buccal mucosa cells, using conventional hypoxanthine phosphoribosyltransferase activity functional assays, sequencing of mitochondrial DNA after specific gene amplification, and measurement of GPI-anchored deficient cells in blood and bone marrow. | No | No |
| C.5 | Assays of immune function of T-cells, including intracellular cytokine staining, ELISPOT, semiquantitative gene amplification for gamma-interferon, tumor necrosis factor, interleukin-2, and other cytokines, and functional assessment in co-culture using specific neutralizing monoclonal antibodies. In addition, peripheral blood lymphocytes are subjected to spectratyping for CDR3 size distribution as well as nucleotide sequence of CDR3 peaks obtained. | No | No |
| C.6 | Studies of engraftment of human normal and diseased bone marrow and peripheral blood in immunodeficient mice in order to determine the presence of hematopoietic repopulating stem cells as well as functional differences among selected populations. | No | No |
| C <b>.7</b> | Flow cytometric analysis of blood and bone marrow for lymphocyte phenotype, especially for evidence of activation of lymphocytes, for markers of apoptosis, and for antigens associated with primitive and mature hematopoietic cell populations. | No | No |
| C <b>.8</b> | Flow cytometric analysis of blood and bone marrow for hematopoietic stem cell progenitors and CD34 positive cells. | No | No |
| C. <b>9</b> | Studies of chromosomal instability in myelopdysplastic syndromes including BM cell and CD34 cell response to PAS crosslinking and examination of the cytotoxic effect of lymphocytes to the abnormal clone of cells. | No | No |
| C.10 | Surface Enhanced Laser/Desorption Ionization (SELDI) time-of-flight mass spectrometry (Ciphergen) (proteomics methodology). | No | No |
| C.11 | Mitochondrial DNA (mtDNA) sequence heterogeneity. | No | No |
| C.12 | Measurement of EBV viral load. | No | No |
| C.13 | Measurement of EBV LMP-1 via RT-PCR for LMP-1 RNA or flow cytometry for LMP-1. | No | No |
| C.14 | Outgrowth assay of EBV transformed B cells. | No | No |
| C.15 | Quantification of serumchemokines and cytokines (e.g. SDF-1, IL-10, IL-6, CXCR4, CXCL12). | No | No |

| C.16 | Quantification of EBV cytotoxic T cells (tetramerstaining). | No | No |
|---|---|---|---|
| C.17 | Telomere length measurement by Southern blot, Q-PCR, flow-fish, in situ | No | No |
| C.17 | hybridization and STELA | INO | NO |
| C.18 | Telomere repair complex gene mutations by nucleotide sequencing of some or all of the following: <i>DKC1</i> , <i>TERC</i> , <i>TERT</i> , <i>SBDS</i> , <i>NOp10</i> , <i>NHP2</i> . | No | No |
| C.19 | Analysis of inflammatory markers and/or bacterial, viral, fungal or protozoal elements in plasma or serum using molecular, colorimetric, enzymatic, flow cytometric or other assays in subjects receiving immunosuppressive therapy, chemotherapy and/or bone marrow transplantation. | No | No |
| C.20 | Confocal microscopic imaging of bone marrow. | No | No |
| C.21 | Characterization of intracellular signaling proteins by cell permeabilization and flow cytometry, and quantitative immunoblots. | No | No |
| C.22 | Assays for chromosomal aneuploidy by florescence in situ hybridization (FISH) and other molecular techniques. | No | No |
| C.23 | Conversion of human dermal fibroblasts into hematopoietic progenitors using Oct4 transfection. | No | No |
| D | Virus Discovery Section (Dr. Neal Young) THESE ASSAYS WILL NOT BE PERFORMED ON SAMPLES FROM HEALTHY PEDIATRIC DONORS | | |
| D.1 | Assays of serum, blood cells, and bone marrow cells for B19 parvovirus and possible B19 variants using gene amplification, cell culture, and hematopoietic colony inhibition assays. | No | N/A |
| <b>D.2</b> | Assays of blood, bone marrow, liver, and other tissues for potentially novel viruses, using a variety of techniques including RNA and DNA assays, differential display, gene amplification with conserved and random primers, cell culture assays, immunohistochemical methods, and inocculation of mice, rabbits, and monkeys, as well as antibody measurements. | No | N/A |
| D.3 | Assays of blood, bone marrow, and liver for known viruses, including herpesviruses such as cytomegalovirus, human herpesviruses 6, 7, and 8, enteric viruses such as A-6, circiviruses, and parvoviruses, using assays as in (2). | No | N/A |
| D.4 | Spectra-typing of blood cells to determine response to known or putative viral infections. | No | N/A |
| D.5 | HLA typing or subtyping to determine risk factors/determinants for hepatitis-AA studies. | No | N/A |
| D.6 | Cytotoxic lymphocyte assays with intracellular cytokine measurement for determining anti-viral response and lymphocyte cloning to obtain clones with specific antiviral activity. | No | N/A |
| E | Solid Tumor Section (Dr. Richard Childs) | | |
| E.1 | Cr51 cytotoxicity assay to evaluating killing of patient tumor cells by patient NK cell clones and T-cells. | No | No |
| E.2 | ELISA for IL-12 maturity of DC's made from subjects monocytes. | No | No |
| E.3 | ELISA for IFN ã to evaluate specificity of CTL clones. | No | No |
| E.4 | H thymidine uptake to evaluate proliferation potential of antigen specific T-cells. | No | No |
| E.5 | PCR of STR to assess chimerism status of cellular subsets grown in-vitro or retrieved from subjects post-transplant. | No | No |
| E.6 | Flow sorting of PBL and/or tissue samples to evaluate chimerism of different subsets. | No | No |
| E.7 | Surface marker analysis of peripheral blood mononuclear cells using flow cytometry. | No | No |
| 1 | cDNA expression arrays to evaluate T-cells expression/gene patterns in subjects with | <b>N</b> T | No |
| E.8 | GVHD and a GVT effect. | No | No |

| E.10 | VHL mutation analysis on kidney cancer tissue. | No | No |
|---|---|---|---|
| E.11 | Transduction of dendritic and tissue cells with tumor antigens using plasmids, viral vectors and hybrid fusions. | No | No |
| E.12 | Lasar capture microdisection of cells from tumor biopsies and tissue samples to determine origin (donor vs patient). | No | No |
| E.13 | Quantification of polyoma virus BK exposure by serology and PCR in stem cell transplant donors and recipients from blood and urine samples. | No | No |
| E.14 | Quantification of polyoma virus BK specific T cells in stem cell transplant donors and recipients from peripheral blood samples. | No | No |
| E.15 | Determination of origin of neovasculature endothelial cells in tumor and tissue samples obtained from subjects post transplant. | No | No |
| E.16 | Quantification of lymphocyte subsets CD34 progenitors and endovasculator progenitors in G-CSF mobilized peripheral cell allografts. | No | No |
| E.17 | Testing for polyoma virus BK latency in CD34 progenitors, B cells and T cells in the G-CSF mobilized peripheral cell allografts. | No | No |
| E.18 | Determination of etiology of membraneous nephropathy using serum from subjects. | No | No |
| E.19 | Serum Proteomic patterns analysis to diagnose complications related to allogeneic transplantation. | No | No |
| E.20 | Determine cell origin (donor vs patient) of tissue samples using IHC, IF, sorting, and FISH. | No | No |
| т. | | | |
| F | Lymphoid Malignancies Section (Dr. Adrian Wiestner) | | |
| F.1 | Culture of cells from research subjects to investigate molecular disease mechanisms, model host tumor interactions, and to test effect of drugs on cell survival and cellular functions. | No | No |
| F.2 | Generation of stable cell lines for the study of hematologic malignancies. | No | No |
| F.3 | Modifications of cells using standard expression systems or biologic molecules, e.g. interfering RNA, to investigate the effects of candidate genes on cellular functions. | | |
| F.4 | Identification and monitoring of B or T cell populations as identified by flow cytometry and by their B cell or T cell receptor expression. | No | No |
| F.5 | Measurement of gene expression in cells or tissues. Techniques frequently used include gene expression profiling on microarrays, quantitative RT-PCR, Western blotting, flow cytometry and ELISA assays. | No | No |
| F.6 | Analysis of chromosomal abnormalities or mutations in malignant cells and non-malignant cells including FISH technology and DNA sequencing. | No | No |
| F.7 | Assays of immune function of B-cells and T-cells, including intracellular cytokine staining, ELISPOT, quantitative RT-PCR for cytokines or other immune regulatory genes. | No | No |
| F.8 | Analysis of antibody specificities in serum and antigen specificity of the B-cell receptor on cells. Techniques may include expression of antibodies in phage display systems, generation of antibodies in cell culture systems and use of such antibodies to screen for cognate antigens. | No | No |
| F.9 | Transplantation of human cells into mice (xenograft model) to study disease biology and to investigate the effect of experimental therapy. | No | No |
| F.10 | Measurements of drug concentrations, biologic molecules and disease markers in | No | No |

#### **APPENDIX C: DEFINITIONS**

ACE inhibitors: Ace inhibitors may increase the nephrotoxicity of cyclosporine; monitor.

Allopurinol: Allopurinol may increase the levels/effects of cyclosporine; monitor cyclosporine concentrations.

Amiodarone: Amiodarone may increase the levels/effects of cyclosporine; monitor cyclosporine concentrations.

Androgens: Androgens may increase the levels/effects of cyclosporine; monitor cyclosporine concentration and for signs/symptoms of renal and/or hepatic toxicity (seen with danazol, fluoxymesterone, methyltestosterone, nandrolone, oxandrolone, oxymetholone, stanozolol, testolactone, and testosterone).

Antacids: Antacids may decrease the levels/effects of cyclosporine.

Antibiotics: Concomitant use may potentiate renal dysfunction (seen with ciprofloxacin, gentamicin, tobramycin, vancomycin, trimethoprim and sulfamethoxazole); increased cyclosporine concentrations by inhibiting cyclosporine metabolism (seen with azithromycin, clarithromycin, erythromycin, and norfloxacin, quinupristin/dalfopristin); may decrease cyclosporine concentrations by inducing cyclosporine metabolism (seen with nafcillin, and rifampin); may decrease immunosuppressant effects (seen with ciprofloxacin); CNS disturbances, seizures (seen with imipenem); imipenem may increase the levels/effects of cyclosporine (monitor for neurotoxicity).

Anticonvulsants: Anticonvulsants may decrease the levels/effects of cyclosporine (seen with carbamazepine, oxcarbazepine, phenobarbital, and phenytoin); monitor cyclosporine concentrations.

Antifungals: Concomitant use may potentiate renal dysfunction (seen with amphotericin B, ketoconazole). May increase cyclosporine concentrations by inhibiting cyclosporine metabolism (seen with fluconazole, itraconazole, ketoconazole, and voriconazole); monitor serum concentrations and renal function.

Antimalarials: Antimalarials may increase the levels/effects of cyclosporine; monitor (seen with chloroquine, hydroxychloroquine, primaquine).

Antineoplastics: Antineoplastics may increase the levels/effects of cyclosporine; monitor for renal dysfunction (seen with melphalan). Cyclosporine may increase the levels/effects of antineoplastics (seen with doxorubicin, etoposide and etoposide phosphate); consider reducing the dose of etoposide and etoposide phosphate by 50% with concomitant administration.

Bosentan: Cyclosporine may increase the levels/effects of bosentan. Bosentan may decrease the levels/effects of cyclosporine. Concurrent use is contraindicated.

Bromocriptine: Increases cyclosporine concentrations by inhibiting cyclosporine metabolism

Calcium channel blockers (eg, diltiazem, nicardipine, verapamil): Calcium channel blockers may increase the levels/effects of cyclosporine; monitor cyclosporine concentrations. Nifedipine has been reported to increase the risk of gingival hyperplasia.

11-H-0064 Am L


Carbonic anhydrase inhibitors: Carbonic anhydrase inhibitors may increase the levels/effects of cyclosporine (seen with acetazolamide, dichlorphenamide, methazolamide; exceptions are brinzolamide, dorzolamide); monitor.

Caspofungin: Cyclosporine may increase the levels/effects of caspofungin; monitor for hepatotoxicity.

Colchicine: Colchicine may increase the levels/effects of cyclosporine; monitor for nephrotoxicity. Cyclosporine may

increase levels/effects of colchicine; monitor for hepatotoxicity and myopathies.

Corticosteroids: Systemic corticosteroids may increase the levels/effects of cyclosporine (reported with methylprednisolone). Cyclosporine may increase the levels/effects of systemic corticosteroids. Convulsions have

been reported with high-dose methylprednisolone.

CYP3A4 inducers: CYP3A4 inducers may decrease the levels/effects of cyclosporine. Example inducers include aminoglutethimide, carbamazepine, nafcillin, nevirapine, oxcarbazepine, phenobarbital, phenytoin, and

rifamycins.

CYP3A4 inhibitors: May increase the levels/effects of cyclosporine. Example inhibitors include azole antifungals,

clarithromycin, diclofenac, doxycycline, erythromycin, imatinib, isoniazid, nefazodone, nicardipine, propofol,

protease inhibitors, quinidine, telithromycin, and verapamil.

CYP3A4 substrates: Cyclosporine may increase the levels/effects of CYP3A4 substrates. Example substrates include

benzodiazepines, calcium channel blockers, cyclosporine, mirtazapine, nateglinide, nefazodone, sildenafil (and

other PDE-5 inhibitors), tacrolimus, and venlafaxine. Selected benzodiazepines (midazolam and triazolam),

cisapride, ergot alkaloids, selected HMG-CoA reductase inhibitors (lovastatin and simvastatin), and pimozide are

generally contraindicated with strong CYP3A4 inhibitors.

Digoxin: Cyclosporine may increase the levels/effects of digoxin; severe digitalis toxicity has been observed.

Estrogen derivatives: Estrogen derivatives may increase the levels/effects of cyclosporine; monitor cyclosporine

concentrations and for signs/symptoms of hepatotoxicity.

Ezetimibe: Ezetimibe may increase the levels/effects of cyclosporine. Cyclosporine may increase the levels/effects of

ezetimibe.

Griseofulvin: Griseofulvin may decrease the levels/effects of cyclosporine.

H<sub>2</sub> blockers: H<sub>2</sub> blockers may increase the levels/effects of cyclosporine; monitor cyclosporine concentrations (seen

with cimetidine, famotidine, ranitidine).

HMG-CoA reductase inhibitors: Cyclosporine may increase levels/effects of HMG-CoA reductase inhibitors,

resulting in myalgias, rhabdomyolysis, acute renal failure; dosage adjustments of HMG-CoA reductase inhibitors

are recommended.

Imatinib: May increase cyclosporine serum concentrations by inhibiting cyclosporine metabolism; monitor.

Metoclopramide: Metoclopramide may increase the levels/effects of cyclosporine.

11-H-0064 Am L


Methotrexate: May increase cyclosporine concentrations and toxicity. Cyclosporine may increase the levels/effects of methotrexate and decreases plasma levels of its metabolite; monitor closely for signs of methrotrexate toxicity.

Minoxidil: Cyclosporine may increase the adverse/toxic effects of minoxidil; may lead to severe hypertrichosis.

NSAIDs: May increase the levels/effects of cyclosporine; concomitant use may potentiate renal dysfunction, especially in dehydrated patients (seen with diclofenac, naproxen, sulindac). Cyclosporine may increase levels/effects of diclofenac; the lowest possible dose of diclofenac should be used

Octreotide: Octreotide may decrease the levels/effects of cyclosporine; monitor cyclosporine concentrations.

Orlistat: Orlistat may decrease the levels/effects of cyclosporine; orlistat may decrease the absorption of oral cyclosporine formulations.

Pimecrolimus: Cyclosporine may increase serum levels/effects of pimecrolimus; monitor.

Probucol: Probucol may decrease the levels/effects of cyclosporine; monitor.

Progestins: Progestins may increase the levels/effects of cyclosporine; monitor for hepatotoxicity.

Protease inhibitors: Formal interaction studies have not been done; protease inhibitors are known to inhibit CYP3A4 and may increase the levels/effects of cyclosporine; use caution when using cyclosporine with indinavir, nelfinavir, ritonavir, or saquinavir.

Repaglinide: Cyclosporine may increase levels/effects of repaglinide; monitor.

Rifamycin derivatives (rifabutin, rifampin, rifapentine): May increase the metabolism, via CYP isoenzymes, of cyclosporine.

Sirolimus: Cyclosporine may increase serum levels/effects of sirolimus. Sirolimus may increase the adverse/toxic effects of cyclosporine. Concurrent therapy may increase the risk of HUS/TTP/TMA. Administer sirolimus 4 hours after cyclosporine to minimize the increase in sirolimus blood levels. Interaction may also occur with concomitant administration of temsirolimus (a pro-drug of sirolimus),

Sitaxsentan [CAN]: Cyclosporine may increase the levels/effects of sitaxsentan; concurrent use is contraindicated.

Sulfasalazine: Sulfasalazine may decrease the levels/effects of cyclosporine.

Sulfinpyrazone: Sulfinpyrazone may decrease the levels/effects of cyclosporine; monitor.

Ticlopidine: Ticlopidine may decrease the levels/effects of cyclosporine.

Vaccines: Vaccination may be less effective; avoid use of live vaccines during therapy.

11-H-0064 Am L
